CLINICAL TRIAL: NCT02820844
Title: A Phase III Study to Evaluate the Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Patients With Overactive Bladder
Brief Title: Efficacy and Safety of GSK1358820 in Subjects With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204947
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder; Botulinum toxin type A; Urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Anti-Infective Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1358820 Injection 100 U (Experimental): Initially, subjects will receive a single (double-blind) treatment with GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia. If the criteria for re-treatment are met between 12 and 36 weeks after the first treatment, subjects will receive a second treatment with GSK1358820 (open-label). A third treatment with GSK1358820 (open-label) may be given until 36 weeks after the first treatment, upon meeting the criteria, provided a minimum of 12 weeks elapse since previous treatment.
  Subjects will receive prophylactic antibiotic therapy beginning up to 3 days prior to treatment and continuing up to 3 days following treatment.
  Interventions: Drug: GSK1358820; Drug: Antibiotic therapy; Other: Bladder diary; Other: King's Health Questionnaire (KHQ); Other: Overactive Bladder Symptom Score (OABSS); Other: Treatment Benefit Scale (TBS)
- Placebo Injection (Placebo Comparator): Initially, subjects will receive a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia. If the criteria for re-treatment are met between 12 and 36 weeks after the first treatment, subjects will receive a second treatment, this time with open-label GSK1358820. A third treatment with open-label GSK1358820 may be given until 36 weeks after the first treatment, upon meeting the criteria, provided a minimum of 12 weeks elapse since previous treatment.
  Subjects will receive prophylactic antibiotic therapy beginning up to 3 days prior to treatment and continuing up to 3 days following treatment.
  Interventions: Drug: GSK1358820; Drug: Placebo; Drug: Antibiotic therapy; Other: Bladder diary; Other: King's Health Questionnaire (KHQ); Other: Overactive Bladder Symptom Score (OABSS); Other: Treatment Benefit Scale (TBS)

INTERVENTIONS:
Drug: GSK1358820 — GSK1358820 injection contains botulinum toxin type A (100 U), sodium chloride (0.9 milligrams [mg]), and human serum albumin (0.5 mg). 10 mL of the drug will be injected at 20 sites (0.5 mL at each site) in the detrusor muscle, spaced approximately 1 centimeter (cm) apart. The injection will be administered under local anesthesia, via cystoscopy. Permitted anesthesia options for cystoscopy are intraurethral lidocaine (or similar) gel, and for treatment administration, installation of 1-2% lidocaine (or similar anesthetic) into the bladder.
Drug: Placebo — Placebo injection is made up of sodium chloride (0.9 mg). 10 mL of the injection will be injected at 20 sites (0.5 mL at each site) in the detrusor muscle, spaced approximately 1 cm apart. The injection will be administered under local anesthesia, via cystoscopy. Permitted anesthesia options for cystoscopy are intraurethral lidocaine (or similar) gel, and for treatment administration, installation of 1-2% lidocaine (or similar anesthetic) into the bladder.
  Arms: Placebo Injection
Drug: Antibiotic therapy — Subjects will use prophylactic antibiotic therapy approved for the indication of UTIs, at the discretion of the investigator, with the exception of those in the class of aminoglycosides. The therapy will begin 1 to 3 days prior to the administration of study treatment, and continue for 1 to 3 days following the treatment.
Other: Bladder diary — The bladder diary is a self-reporting tool to record subject's data on micturition. Subjects will enter data in the diary over 3 consecutive days. During Screening, data will be collected within 28 days prior to first treatment. During treatment periods, data will be collected within a week prior to each scheduled visit. The bladder diary will capture the following information: 1) Date and time of urinary episode, 2) episodes of micturition, 3) episodes of urinary incontinence, 4) episodes of urgency, 5) intensity of urgency, 6) episodes of nocturia, 7) use of CIC, and 8) urine volume. Diary data will not be collected when a subject experiences symptoms of a UTI.
Other: King's Health Questionnaire (KHQ) — The KHQ will assess the impact of urinary incontinence on QOL. It is a questionnaire with 21 items and the following 9 domains: 1) General health, 2) Incontinence impact, 3) Role limitations, 4) Physical limitations, 5) Social limitations, 6) Personal relationships, 7) Emotion, 8) Sleep/energy, 9) Severity measure. The items are answered by subjects themselves, and scores are summated using a defined algorithm.
Other: Overactive Bladder Symptom Score (OABSS) — The OABSS will comprehensively assess symptoms of OAB, such as frequency of micturition, nocturia, urinary urgency, and urge incontinence. It consists of 4 questions which will be responded by subjects themselves, by selecting the most appropriate answer for each question.
Other: Treatment Benefit Scale (TBS) — The TBS consists of one question ("My condition has"), to which the subject will answer by selecting one of the following responses: greatly improved, improved, not changed, worsened. The TBS will assess treatment benefit of GSK1358820.

SUMMARY:
GSK1358820 is a botulinum neurotoxin A complex that has been approved for the treatment of overactive bladder (OAB) in several countries, however, it has not been approved for OAB treatment in Japan. This study has been planned to evaluate the efficacy and safety of GSK1358820 in Japanese OAB patients with urinary incontinence whose symptoms have not been adequately managed with other medications for OAB.

The primary objective of this study is to evaluate the superiority of a single dose treatment of GSK1358820 100 units (U) compared with placebo.

The study comprises a screening phase up to 28 days, followed by a double-blind treatment phase of 12 to 48 weeks wherein subjects will receive a single treatment of either GSK1358820 100 U injection or Placebo injection, in a ratio of 1:1, with further stratification within the treatment arms according to the number of urinary urge incontinence episodes during screening. Subjects meeting the criteria for re-treatment will receive a second and third treatment. Each re-treatment will be with open-label GSK1358820 100 U injection, and will be spaced at least 12 weeks from the previous treatment.

The total duration of participation for any subject will not exceed 52 weeks, including screening and the 48-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=20 years at the time of signing the informed consent.
* Subject has symptoms of OAB (frequency and urgency) with urinary incontinence for a period of at least 6 months immediately prior to screening, determined by documented subject history.
* Subject has not been adequately managed with one or more medications (that is, anticholinergics or beta-3 adrenergic receptor agonist) for treatment of their OAB symptom. 'Not adequately managed' is defined as: An inadequate response after at least a 4-week period of OAB medication(s) on an approved optimized dose(s), that is, subject is still incontinent despite medication(s) for OAB; or limiting side effects (that is, condition that subject reduced dosage or discontinued the medication due to side effect after at least a 2-week period of OAB medication(s) on an approved optimized dose(s)).
* Subject who experiences all of the following, in the 3-day subject bladder diary completed during the screening phase:

  1. >= 3 episodes of urinary urgency incontinence, with no more than one urgency incontinence-free day
  2. urinary frequency (defined as an average of >= 8 micturitions [toilet voids] per day, that is, a total of >= 24 micturitions)
* Subject is willing to use clean intermittent catheterization (CIC) to drain urine if it is determined to be necessary by the investigator (or subinvestigator).
* Body weight >=40 kilograms (kg) at screening.
* Males or females:

  1. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until the study exit:

     * Vasectomy with documentation of azoospermia.
     * Male condom plus partner use of one of the contraceptive options below: Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; or oral contraceptive, either combined or progestogen alone.

     These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
  2. Female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine or serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

     • Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

     Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

     • Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until the study exit. This list of highly effective methods (approved in Japan) is provided below, and it does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis: Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

     These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Subject has given signed informed consent, including compliance with the requirements and restrictions listed in the consent form and in this protocol (example, using the toilet without assistance, complete bladder diaries and questionnaires, is able to collect volume voided per micturition measurements over a 24-hour period, and attend all study visits in the opinion of the investigator (or subinvestigator).

Exclusion Criteria:

* Subject has symptoms of OAB due to any known neurological reason (example, spinal cord injury, multiple sclerosis, cerebrovascular accident, Alzheimer's disease, Parkinson's disease, etc.)
* Subject has a predominance of stress incontinence determined by subject history.
* Subject has a history or evidence of any diseases, functional abnormalities or bladder surgery, other than OAB, that may have affected bladder function including but not limited to:

  1. Bladder stones (including bladder stone surgery) within 6 months prior to screening or confirmed occurrence of bladder stones at the screening phase
  2. Surgery (including minimally invasive surgery) within 1 year of screening for stress incontinence or pelvic organ prolapse
  3. Current use of an electrostimulation/neuromodulation device for treatment of urinary incontinence. Note: Use of any implantable device is prohibited within 4 weeks prior to initiation of screening phase and throughout the study period. Use of any external device is prohibited within 7 days prior to the start of the screening phase
  4. History of interstitial cystitis, in the opinion of the investigator (or subinvestigator)
  5. Past or current evidence of hematuria due to urological/renal pathology or uninvestigated hematuria. Subjects with investigated hematuria may enter the study if urological/renal pathology has been ruled out to the satisfaction by the investigator (or subinvestigator).
  6. Past or current history of bladder cancer or other urothelial malignancy, positive result of urine cytology or uninvestigated suspicious urine cytology results at the Screening phase. Suspicious urine cytology abnormalities require that bladder cancer or other urothelial malignancy has been ruled out to the satisfaction of the investigator according to local site practice.
  7. An active genital infection, other than genital warts, either concurrently or within 4 weeks prior to Screening
  8. Male with previous or current diagnosis of prostate cancer or a prostate specific antigen (PSA) level of >10 nanograms (ng)/mL at Screening. Subjects with a PSA level of >= 4 ng/mL but <= 10 ng/mL must have prostate cancer ruled out to the satisfaction of the investigator (or subinvestigator) according to local site practice.
  9. Evidence of urethral and/or bladder outlet obstruction, in the opinion of the investigator (or subinvestigator)
* Subject has a history of 2 or more urinary tract infections (UTIs) within 6 months of initiation of Treatment phase 1 (Week 0) or current administration of prophylactic antibiotics to prevent chronic UTIs
* Subject has a positive urine dipstick reagent strip test at initiation of Treatment phase 1 (Week 0) for nitrites or leukocyte esterase, or who are considered by the investigator (or subinvestigator) to have UTI.
* Subject has a serum creatinine level >2 times the upper limit of normal (ULN) at screening.
* Alanine aminotransferase (ALT) > 2xULN; and bilirubin > 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Subject has current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Notes:

  1. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice, or cirrhosis
  2. Chronic stable hepatitis B and C (example, presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody [HCVAb] test result within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria
* QT corrected (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block from the result of electrocardiogram (ECG) at screening. Notes:

  1. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read
  2. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial
* Subject has hemophilia or other clotting factor deficiencies or disorders that cause bleeding diathesis.
* Subject received anticholinergic, beta-3 adrenergic receptor agonist or any other medications or therapies to treat symptoms of OAB, including nocturia, within 7 days prior to the start of the screening phase.
* Subject has been treated with any intravesical pharmacologic agent (example, capsaicin, resiniferatoxin) for OAB symptoms within 12 months prior to initiation of Treatment phase 1 (Week 0).
* Subject has previous or current use of botulinum toxin therapy of any serotype for the treatment of any urological condition.
* Subject has previous use within 12 weeks prior to initiation of Treatment phase 1 (Week 0) or current use of botulinum toxin therapy of any serotype for any non-urological condition or beauty care.
* Subject has been immunized for botulinum toxin of any serotype.
* Subject cannot withhold any antiplatelet or anticoagulant therapy or medications with anticoagulative effects for 3 days prior to initiation of Treatment phase 1 (Week 0). Some medications may need to be withheld for >3 days, per clinical judgment of the investigator (or subinvestigator).
* Subject has not initiated appropriate antibiotic medication 1 to 3 days prior to the initiation of Treatment phase 1 (Week 0).
* Subject uses CIC or indwelling catheter to manage their urinary incontinence.
* Subject has a history of sensitivity to any of the study medications, medications used in the study (including anesthesia), or their components or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Subject has any medical condition that may put them at increased risk with exposure to GSK1358820 including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis.
* Females who are pregnant, nursing or planning a pregnancy during the study.
* Subject has a PVR urine volume of >100 mL at screening phase. The PVR measurement can be repeated once; the subject is to be excluded if the repeated measure is above 100 mL.
* Subject has had urinary retention or an elevated PVR urine volume within 6 months of screening that has been treated with an intervention (such as catheterization). Voiding difficulties as a result of surgical procedures that resolved within 24 hours are not exclusionary.
* Subject has a 24-hour total volume of urine voided >3000 mL of urine collected over 24 consecutive hours during the 3-day bladder diary collection period in the Screening phase.
* Subject is currently participating in or has previously participated in another therapeutic study within 30 days prior to the start of the Screening phase.
* Subject has any condition or situation which, in the investigator's (or subinvestigator's) opinion, puts the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Japan (25):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20738

REFERENCES:
- [Background] Yokoyama O, Honda M, Yamanishi T, Sekiguchi Y, Fujii K, Nakayama T, Mogi T. OnabotulinumtoxinA (botulinum toxin type A) for the treatment of Japanese patients with overactive bladder and urinary incontinence: Results of single-dose treatment from a phase III, randomized, double-blind, placebo-controlled trial (interim analysis). Int J Urol. 2020 Mar;27(3):227-234. doi: 10.1111/iju.14176. Epub 2020 Jan 20. PMID 31957922
- [Derived] Yokoyama O, Honda M, Yamanishi T, Sekiguchi Y, Fujii K, Kinoshita K, Nakayama T, Ueno A, Mogi T. Efficacy and safety of onabotulinumtoxinA in patients with overactive bladder: subgroup analyses by sex and by serum prostate-specific antigen levels in men from a randomized controlled trial. Int Urol Nephrol. 2021 Nov;53(11):2243-2250. doi: 10.1007/s11255-021-02962-z. Epub 2021 Jul 22. PMID 34292493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of GSK1358820 (botulinum toxin type A) in participants with overactive bladder. This was a multicenter study conducted in Japan.
Pre-assignment Details: A total 354 participants were screened, of which, 104 failed screening and 250 were randomized. Of the 250 randomized, 248 received GSK1358820 100 units (U) or placebo. One participant did not receive treatment due to defective investigational product vial and the other participant was met with protocol exclusion criteria before dosing.
Groups:
- Treatment Cycle 1: Placebo: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1).
- Treatment Cycle 1: GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1).
- Treatment Cycle 2: Placebo / GSK1358820 100 U: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received GSK1358820 100 U in the open-label Treatment Phase 2 (Treatment Cycle 2).
- Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 (Treatment Cycle 2).
- Treatment Cycle 3: Placebo / GSK1358820 100 U: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received GSK1358820 100 U in the open-label Treatment Phase 2 (Treatment Cycle 2) and further received re-treatment with GSK1358820 100 U in Treatment Phase 2 (Treatment Cycle 3).
- Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 (Treatment Cycle 2) and further re-treatment with GSK1358820 100 U in Treatment Phase 2 (Treatment Cycle 3).
Period: Double-blinded (Up to 48 Weeks)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Started | 124 | 124 | 0 | 0 | 0 | 0
Completed | 119 | 115 | 0 | 0 | 0 | 0
Not Completed | 5 | 9 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Reached stopping criteria | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-label(2nd Treatment-Up to 48 Weeks)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Started | 0 | 0 | 108 | 88 | 0 | 0
Completed | 0 | 0 | 99 | 84 | 0 | 0
Not Completed | 0 | 0 | 9 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 2 | 0 | 0
Period: Open-label(3rd Treatment-Up to 48 Weeks)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Started | 0 | 0 | 0 | 0 | 56 | 43
Completed | 0 | 0 | 0 | 0 | 54 | 42
Not Completed | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Reached stopping criteria | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 milliliter [mL] each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1. Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment could receive re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 until Week 36 after the first treatment and up to 2 times with an interval of at least 12 weeks between treatments.
- GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1. Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment could receive re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 until Week 36 after the first treatment and up to 2 times with an interval of at least 12 weeks between treatments.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1358820 100 U | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (12.19) | 65.6 (12.43) | 65.9 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 186
  Male | 30 | 32 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese Heritage | 124 | 124 | 248

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes at Week 12 After the First Treatment
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1), excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes were calculated using formula; number of "Yes" response to the diary question of accidental urinary leakage divided by number of valid diary days in the visit. Baseline is the latest pre-dose 3- day diary assessment which has at least one valid diary day. Change from Baseline is any visit value minus Baseline value. Adjusted mean and standard error of adjusted mean has been reported.
Time Frame: Baseline (Pre-dose on Day 1) and Week 12 in Treatment Cycle 1
Population: Full Analysis Set 1(FAS1) Population comprised of all randomized participants who had at least 1 post-Baseline efficacy assessment. Only those participants with data available at specified time point were analyzed.
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 122 | 122
Episodes | -1.25 (0.375) | -3.42 (0.381)
Statistical Analysis 1: Comparison: Treatment Cycle 1: Placebo vs Treatment Cycle 1: GSK1358820 100 U; Test type: Other; p < 0.001, MMRM — Analysis was performed using mixed-model for repeated measures (MMRM) with treatment, site, visit, treatment-by-visit interaction, Baseline value, Baseline-by-visit interaction as fixed effects; Mean Difference (Net) = -2.16, 95% CI 2-sided [-3.14 to -1.18] — Mean difference (Net) at Week 12 has been presented

2. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in the Average Volume Voided Per Micturition at Week 12 After the First Treatment
Description: The total volume voided was measured and recorded by participants in the bladder diary, over a 24-hour period during the 3-day diary collection period. Volume voided per micturition was determined by dividing the total urine volume collected in 24-hour period by the participants with the number of the urinary volume records which are not missing. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value. Adjusted mean and standard error of adjusted mean has been reported.
Time Frame: Baseline (Pre-dose on Day 1) and Week 12 in Treatment Cycle 1
Population: FAS1 Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (Standard Error); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 122 | 122
Milliliter | -0.22 (4.329) | 29.47 (4.390)
Statistical Analysis 1: Comparison: Treatment Cycle 1: Placebo vs Treatment Cycle 1: GSK1358820 100 U; Test type: Other; p < 0.001, MMRM — Analysis performed using MMRM, with treatment, site, visit, Baseline urinary urgency incontinence (UUI) episodes over 3 day diary (<=9 or >=10), treatment-by-visit interaction, Baseline value, Baseline-by-visit interaction as fixed effects; Mean Difference (Net) = 29.69, 95% CI 2-sided [18.47 to 40.91] — Mean difference (Net) at Week 12 has been presented

3. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Changes From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1), excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage with number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42 and Week 48 in Treatment Cycle 1
Population: FAS1 Population. All the participants in this population were analyzed (124, 124 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.84 (2.883) | -3.24 (4.355)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -0.83 (3.022) | -3.62 (4.447)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.92 (3.402) | -3.41 (4.394)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -1.22 (3.422) | -4.07 (3.477)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -2.51 (1.704) | -3.88 (3.516)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -2.52 (1.920) | -3.05 (3.826)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -2.03 (2.153) | -3.27 (2.508)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -2.03 (2.079) | -3.42 (3.022)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -1.73 (2.732) | -3.07 (3.037)

4. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Changes From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1), excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage with number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value. FAS2 Population comprised all randomized participants who had at least 1 post-2nd treatment efficacy assessment after 2nd treatment.
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, and Week 36 in Treatment Cycle 2
Population: FAS2 Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Episodes
Groups:
- Treatment Cycle 2: Placebo / GSK1358820 100 U: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received GSK1358820 100 U in Treatment Phase 2 (Treatment Cycle 2).
- Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 (Treatment Cycle 2) until Week 36 after the first treatment.
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.54 (3.645) | -2.86 (4.091)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -4.34 (3.880) | -4.61 (3.610)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -3.92 (3.760) | -4.44 (3.860)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -3.77 (3.776) | -4.49 (4.123)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -3.75 (3.639) | -4.21 (3.776)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -3.93 (4.202) | -5.22 (3.370)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -3.91 (4.366) | -4.58 (3.967)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -4.63 (4.142) | -2.78 (3.060)

5. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Changes From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1), excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage with number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value. FAS3 Population comprised of all randomized participants who had at least 1 post-3rd treatment efficacy assessment after 3rd treatment.
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Episodes
Groups:
- Treatment Cycle 3: Placebo / GSK1358820 100 U: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received GSK1358820 100 U in Treatment Phase 2 (Treatment Cycle 3).
- Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U: Participants received a single (double-blind) dose of GSK1358820 (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 100 U (open-label) in Treatment Phase 2 (Treatment Cycle 3) until Week 36 after the first treatment.
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -2.99 (3.476) | -3.92 (4.376)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -3.53 (4.370) | -4.57 (4.684)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -3.43 (3.952) | -5.10 (4.689)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -3.50 (3.664) | -4.60 (4.504)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -3.09 (4.306) | -3.80 (5.103)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -2.00 (1.886) | -0.83 (1.232)

6. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Change From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1), excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes was calculated from bladder diary data recorded by the participants during the 3-day diary collection period by dividing the number of 'Yes' response to the diary question of accidental urinary leakage with number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -12.68 (45.315) | -33.38 (202.484)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -7.97 (74.450) | -38.84 (201.345)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -8.82 (61.933) | -38.27 (146.283)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -13.19 (140.232) | -64.41 (37.980)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -58.96 (46.668) | -69.46 (38.644)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -64.58 (47.877) | -47.52 (60.743)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -61.62 (44.722) | -62.82 (39.971)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -48.59 (62.571) | -63.46 (46.638)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -34.51 (91.409) | -63.06 (36.960)

7. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Change From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 6
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30 and Week 36 in Treatment Cycle 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=108,88 | 6.68 (82.009) | -29.45 (51.218)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -67.19 (45.799) | -65.02 (34.778)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -65.64 (42.063) | -61.88 (43.428)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -62.41 (45.304) | -57.43 (45.561)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -58.48 (38.500) | -59.90 (47.789)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -62.54 (53.503) | -79.20 (24.398)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -62.58 (46.592) | -72.34 (29.508)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -71.28 (33.179) | -65.09 (42.285)

8. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Change From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 6
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=56,43 | -37.29 (46.169) | -41.20 (30.656)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -48.51 (63.535) | -54.46 (44.164)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -52.66 (54.383) | -60.40 (35.855)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -53.49 (43.246) | -54.62 (33.369)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -39.80 (45.118) | -44.10 (43.035)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -16.85 (14.397) | -29.06 (37.514)

9. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: The daily average number of urge incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage and sudden/ urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.64 (2.709) | -3.17 (4.182)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -0.66 (2.939) | -3.44 (4.274)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.69 (3.228) | -3.12 (4.301)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -1.43 (2.587) | -3.78 (3.272)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -2.43 (1.686) | -3.65 (3.220)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -2.50 (1.903) | -2.99 (3.659)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -2.28 (1.650) | -3.09 (2.398)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -2.36 (1.900) | -3.42 (2.951)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -2.27 (1.965) | -3.05 (2.885)

10. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: as for outcome 9
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.36 (3.326) | -2.65 (4.075)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -4.01 (3.529) | -4.41 (3.560)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -3.67 (3.301) | -4.21 (3.733)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -3.46 (3.556) | -4.24 (4.094)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -3.45 (3.238) | -3.88 (3.640)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -3.59 (3.720) | -4.84 (3.359)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -3.65 (3.728) | -4.56 (3.945)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -4.37 (3.169) | -2.78 (3.060)

11. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: as for outcome 9
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -2.69 (3.554) | -3.68 (4.521)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -3.38 (4.221) | -4.37 (4.823)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -3.31 (3.592) | -4.74 (4.946)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -3.31 (3.567) | -4.53 (4.624)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -2.67 (4.505) | -3.59 (5.137)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -2.17 (1.650) | -1.33 (0.609)

12. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: The daily average number of urge incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage and sudden/ urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -12.65 (47.510) | -34.86 (202.832)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -7.81 (75.815) | -40.56 (193.346)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -5.35 (67.599) | -36.86 (143.314)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -30.32 (71.194) | -66.24 (37.732)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -60.58 (47.367) | -72.58 (36.701)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -67.17 (48.289) | -50.68 (60.176)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -66.48 (33.584) | -64.98 (41.020)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -57.05 (59.914) | -72.13 (45.202)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -58.83 (69.302) | -69.56 (35.673)

13. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: as for outcome 12
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=108,88 | 7.31 (67.536) | -27.01 (57.513)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -64.76 (61.700) | -66.40 (35.804)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -66.00 (42.442) | -61.50 (43.730)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -61.39 (49.370) | -55.11 (50.258)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -57.93 (39.299) | -59.27 (48.577)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -59.10 (72.369) | -79.37 (24.927)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -63.64 (51.577) | -72.34 (29.508)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -74.12 (32.549) | -65.09 (42.285)

14. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Change From Baseline in Daily Average Number of Urinary Urgency Incontinence Episodes
Description: as for outcome 12
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=56,43 | -35.51 (47.233) | -35.41 (40.461)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -49.97 (61.305) | -53.60 (53.462)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -54.12 (48.948) | -53.99 (48.401)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -54.34 (44.946) | -55.10 (36.963)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -37.88 (49.474) | -44.81 (45.494)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -18.69 (11.796) | -34.56 (31.169)

15. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Voids
Description: The daily average number of micturition episodes (voids) were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of 'Yes response to the diary question of urination into the toilet with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Voids
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.39 (2.419) | -0.71 (3.363)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -0.26 (2.506) | -1.90 (3.418)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.41 (2.681) | -2.00 (3.447)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -1.00 (3.338) | -2.46 (3.136)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -1.18 (2.703) | -2.34 (3.334)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -1.29 (2.525) | -1.40 (2.895)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -1.39 (2.777) | -2.06 (2.667)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -1.39 (4.044) | -2.06 (2.956)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -0.36 (2.610) | -1.14 (2.453)

16. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Voids
Description: as for outcome 15
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Voids
  Week 0; n=108,88 | -0.16 (2.579) | -1.46 (2.556)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -1.58 (3.473) | -1.68 (3.394)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -2.04 (3.199) | -2.21 (2.879)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -2.22 (3.164) | -1.99 (2.575)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -2.41 (2.312) | -1.53 (2.789)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -2.62 (2.169) | -2.59 (2.738)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -2.48 (3.051) | -2.49 (2.597)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -2.73 (3.037) | -0.39 (3.044)

17. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Voids
Description: as for outcome 15
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Voids
  Week 0; n=56,43 | -1.58 (3.166) | -2.12 (2.495)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -1.57 (3.476) | -2.29 (2.864)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -1.85 (2.917) | -2.62 (2.623)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -1.95 (2.836) | -2.02 (2.173)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -2.12 (3.766) | -1.74 (2.327)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -1.33 (0.943) | -1.08 (0.877)

18. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Change From Baseline in Daily Average Number of Voids
Description: The daily average number of micturition episodes (voids) were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of 'Yes response to the diary question of urination into the toilet with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -1.65 (19.992) | -4.31 (27.295)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -1.05 (20.639) | -12.81 (25.192)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -2.59 (21.271) | -14.12 (25.463)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -4.81 (24.135) | -18.70 (20.675)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -6.21 (18.990) | -18.29 (21.921)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -8.36 (15.789) | -10.35 (21.713)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -8.33 (15.374) | -16.22 (21.705)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -14.26 (38.087) | -15.40 (22.368)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -2.50 (18.160) | -7.82 (22.261)

19. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Change From Baseline in Daily Average Number of Voids
Description: as for outcome 18
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=108,88 | -0.31 (20.076) | -10.14 (18.892)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -11.53 (26.466) | -11.11 (30.081)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -14.87 (23.844) | -16.31 (23.417)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -15.78 (26.649) | -14.52 (20.260)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -19.08 (18.022) | -10.88 (22.318)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -22.08 (16.561) | -18.61 (20.308)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -19.22 (21.626) | -18.90 (20.805)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -19.03 (20.561) | -2.57 (24.843)

20. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Change From Baseline in Daily Average Number of Voids
Description: as for outcome 18
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=56,43 | -9.68 (30.804) | -14.43 (19.179)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -9.81 (30.062) | -15.98 (22.524)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -12.53 (25.204) | -19.34 (20.321)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -13.16 (23.767) | -15.30 (17.431)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -11.60 (32.168) | -13.31 (18.080)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -12.42 (8.142) | -9.07 (5.887)

21. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Average Volume Voided Per Micturition
Description: The total volume voided was measured and recorded by participants in the bladder diary, over a 24-hour period during the 3-day diary collection period. Volume voided per micturition was determined by dividing the total urine volume collected in 24-hour period by the participants with the number of the urinary volume records which are not missing. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Milliliter
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | 3.99 (29.762) | 14.74 (44.121)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | 0.95 (36.800) | 30.19 (52.077)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -1.69 (34.578) | 29.13 (46.480)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | 5.48 (31.328) | 30.67 (49.697)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | 2.37 (36.827) | 31.67 (51.061)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | 6.39 (32.508) | 32.08 (57.263)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | 9.73 (34.867) | 30.34 (44.953)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | 5.34 (31.688) | 17.48 (38.558)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | 6.60 (32.580) | 14.41 (42.699)

22. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 21
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Milliliter
  Week 0; n=108,88 | -2.10 (34.115) | 25.74 (45.213)
  Week 2; n=103,87: number analyzed (Participants) | 103 | 87
  Week 2; n=103,87 | 17.38 (44.216) | 20.44 (51.406)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | 25.80 (50.630) | 29.03 (56.182)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | 26.72 (49.861) | 24.04 (51.918)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | 28.53 (43.876) | 12.34 (50.453)
  Week 24; n=45,20: number analyzed (Participants) | 45 | 20
  Week 24; n=45,20 | 28.88 (50.296) | 22.34 (39.877)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | 38.27 (57.547) | 26.74 (45.696)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | 43.99 (63.155) | 9.49 (69.972)

23. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 21
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Milliliter
  Week 0; n=56,43 | 19.49 (36.341) | 25.60 (35.923)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | 20.32 (38.050) | 25.01 (46.534)
  Week 6; n=53,41: number analyzed (Participants) | 53 | 41
  Week 6; n=53,41 | 28.13 (41.894) | 20.39 (47.654)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | 24.51 (39.670) | 17.33 (45.658)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | 23.51 (56.849) | 18.09 (35.324)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -6.79 (2.180) | 15.57 (45.613)

24. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Change From Baseline in Average Volume Voided Per Micturition
Description: The total volume voided was measured and recorded by participants in the bladder diary, over a 24-hour period during the 3-day diary collection period. Volume voided per micturition was determined by dividing the total urine volume collected in 24-hour period by the participants with the number of the urinary volume records which are not missing. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | 4.47 (24.306) | 14.47 (35.109)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | 3.10 (28.671) | 28.73 (43.846)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | 1.93 (29.197) | 27.42 (41.440)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | 7.61 (27.947) | 28.64 (48.898)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | 6.94 (32.660) | 26.80 (45.728)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | 9.87 (31.384) | 24.39 (36.838)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | 8.51 (24.109) | 26.08 (41.728)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | 8.41 (32.804) | 14.91 (32.231)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | 9.11 (28.104) | 11.98 (36.358)

25. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 24
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=108,88 | 1.72 (28.347) | 24.71 (38.824)
  Week 2; n=103,87: number analyzed (Participants) | 103 | 87
  Week 2; n=103,87 | 16.62 (41.294) | 21.94 (39.385)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | 21.50 (44.146) | 28.51 (43.091)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | 21.92 (41.446) | 23.99 (42.719)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | 25.12 (38.530) | 12.60 (34.000)
  Week 24; n=45,20: number analyzed (Participants) | 45 | 20
  Week 24; n=45,20 | 30.10 (54.874) | 19.48 (30.916)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | 33.02 (69.583) | 20.14 (35.588)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | 39.51 (76.822) | 13.35 (52.100)

26. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 24
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=56,43 | 18.96 (37.442) | 23.41 (33.357)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | 20.24 (37.340) | 25.78 (43.344)
  Week 6; n=53,41: number analyzed (Participants) | 53 | 41
  Week 6; n=53,41 | 25.51 (37.686) | 23.65 (46.594)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | 25.28 (40.894) | 20.05 (40.347)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | 20.23 (45.654) | 19.37 (34.051)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -3.88 (0.051) | 11.46 (36.629)

27. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Urgency Episodes
Description: The daily average number of urgency episodes were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of "Yes" response to the diary question of episode associated with a sudden and urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -1.10 (3.100) | -2.09 (4.826)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -1.39 (3.607) | -3.30 (4.563)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -1.08 (3.809) | -3.39 (4.471)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -2.46 (3.726) | -3.99 (4.173)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -3.47 (3.482) | -4.60 (4.204)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -3.93 (4.172) | -3.78 (5.056)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -3.25 (3.921) | -4.22 (4.514)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -2.88 (4.822) | -4.12 (3.586)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -2.52 (3.659) | -3.57 (3.943)

28. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Urgency Episodes
Description: as for outcome 27
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.79 (3.639) | -2.42 (3.822)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -3.63 (4.580) | -3.69 (4.347)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -4.28 (4.074) | -3.83 (3.962)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -4.10 (4.118) | -3.67 (3.591)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -3.86 (3.972) | -3.06 (3.699)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -4.47 (4.352) | -3.49 (2.662)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -4.06 (5.020) | -3.42 (2.435)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -5.08 (5.582) | -1.72 (4.716)

29. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Urgency Episodes
Description: as for outcome 27
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -2.64 (3.362) | -3.22 (3.668)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -3.28 (4.476) | -3.89 (4.286)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -3.50 (3.878) | -4.40 (4.257)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -3.28 (3.300) | -3.63 (4.093)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -3.14 (4.082) | -2.97 (3.654)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -2.17 (1.650) | -2.00 (2.480)

30. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Change From Baseline in Daily Average Number of Urgency Episodes
Description: The daily average number of urgency episodes were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of "Yes" response to the diary question of episode associated with a sudden and urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -11.62 (36.556) | -12.27 (139.897)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -13.36 (39.284) | -29.25 (99.826)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -6.15 (55.275) | -28.92 (76.618)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -24.56 (67.816) | -41.72 (54.362)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -44.53 (46.229) | -54.05 (45.299)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -45.85 (49.841) | -39.11 (59.666)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -41.35 (47.808) | -49.87 (52.601)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -36.82 (73.233) | -51.54 (44.338)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -35.81 (56.080) | -47.94 (52.200)

31. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Change From Baseline in Daily Average Number of Urgency Episodes
Description: as for outcome 30
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=108,88 | -0.97 (53.493) | -17.59 (52.475)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -34.51 (75.956) | -43.19 (48.933)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -46.94 (41.256) | -42.81 (48.411)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -44.42 (58.087) | -37.61 (44.355)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -41.83 (60.854) | -37.30 (57.929)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -50.30 (62.946) | -50.18 (36.257)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -43.83 (76.751) | -47.11 (35.298)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -42.83 (100.717) | 17.36 (163.104)

32. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Change From Baseline in Daily Average Number of Urgency Episodes
Description: as for outcome 30
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=56,43 | -25.28 (38.080) | -21.29 (56.917)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -31.32 (58.360) | -35.08 (55.559)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -36.80 (45.867) | -36.67 (60.410)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -33.95 (35.729) | -32.80 (62.144)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -28.72 (37.453) | -33.32 (47.860)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -18.69 (11.796) | -18.03 (21.046)

33. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Nocturia Episodes
Description: Nocturia episodes are voids (micturition episodes) that interrupt night sleep. The daily average number of nocturia episodes were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of episodes that awake participants from night sleep with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.09 (0.835) | -0.09 (1.275)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -0.13 (1.091) | -0.26 (1.216)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.03 (1.098) | -0.29 (1.447)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -0.16 (1.247) | -0.53 (1.334)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | 0.04 (1.224) | -0.58 (1.535)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | 0.14 (1.357) | -0.15 (0.825)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | 0.19 (1.453) | -0.21 (1.148)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | 0.30 (1.574) | -0.33 (1.109)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | 0.36 (1.487) | -0.19 (0.940)

34. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Nocturia Episodes
Description: as for outcome 33
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.10 (1.079) | -0.32 (1.303)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -0.32 (1.020) | -0.42 (1.309)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -0.45 (1.079) | -0.45 (1.358)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -0.36 (1.266) | -0.38 (1.331)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -0.33 (1.032) | -0.40 (1.490)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -0.24 (0.831) | -0.03 (0.888)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -0.01 (0.964) | 0.02 (0.831)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | 0.05 (0.987) | 0.61 (1.769)

35. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Nocturia Episodes
Description: as for outcome 33
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -0.44 (1.314) | -0.29 (1.032)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -0.44 (1.410) | -0.31 (1.012)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -0.46 (1.299) | -0.29 (1.070)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -0.72 (1.396) | -0.47 (1.093)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -0.50 (1.212) | -0.34 (1.449)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | 0.33 (0.471) | -0.33 (0.720)

36. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage Changes From Baseline in Daily Average Number of Nocturia Episodes
Description: Nocturia episodes are voids (micturition episodes) that interrupt night sleep. The daily average number of nocturia episodes were calculated from bladder diary data recorded by the participant during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of episodes that awake participants from night sleep with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percent change
  Week 2; n=112, 104: number analyzed (Participants) | 112 | 104
  Week 2; n=112, 104 | -2.92 (78.249) | -0.87 (92.501)
  Week 6; n=112, 102: number analyzed (Participants) | 112 | 102
  Week 6; n=112, 102 | -7.29 (65.866) | -7.81 (86.301)
  Week 12; n=111, 103: number analyzed (Participants) | 111 | 103
  Week 12; n=111, 103 | 7.83 (79.745) | -7.23 (114.564)
  Week 18; n=20, 50: number analyzed (Participants) | 20 | 50
  Week 18; n=20, 50 | 5.01 (142.476) | -29.88 (58.668)
  Week 24; n=15, 41: number analyzed (Participants) | 15 | 41
  Week 24; n=15, 41 | 18.51 (141.097) | -21.27 (97.052)
  Week 30; n=11, 37: number analyzed (Participants) | 11 | 37
  Week 30; n=11, 37 | -3.25 (142.123) | -0.22 (80.388)
  Week 36; n=10, 26: number analyzed (Participants) | 10 | 26
  Week 36; n=10, 26 | 35.52 (206.821) | -8.10 (89.630)
  Week 42; n=9, 22: number analyzed (Participants) | 9 | 22
  Week 42; n=9, 22 | 29.63 (224.354) | -15.72 (94.273)
  Week 48; n=9, 22: number analyzed (Participants) | 9 | 22
  Week 48; n=9, 22 | 38.52 (189.877) | -9.60 (78.016)

37. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage Changes From Baseline in Daily Average Number of Nocturia Episodes
Description: as for outcome 36
Time Frame: as for outcome 7
Population: FAS2 Population. All the participants in this population were analyzed (108, 88 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percent change
  Week 0; n=99,75: number analyzed (Participants) | 99 | 75
  Week 0; n=99,75 | 1.84 (63.835) | -12.98 (68.669)
  Week 2; n=96,74: number analyzed (Participants) | 96 | 74
  Week 2; n=96,74 | -10.92 (68.689) | -19.95 (56.983)
  Week 6; n=97,71: number analyzed (Participants) | 97 | 71
  Week 6; n=97,71 | -19.84 (60.168) | -16.88 (71.816)
  Week 12; n=97,72: number analyzed (Participants) | 97 | 72
  Week 12; n=97,72 | -17.89 (70.405) | -15.74 (65.355)
  Week 18; n=75,39: number analyzed (Participants) | 75 | 39
  Week 18; n=75,39 | -16.10 (68.014) | -12.99 (55.055)
  Week 24; n=38,19: number analyzed (Participants) | 38 | 19
  Week 24; n=38,19 | -17.35 (60.337) | -4.88 (52.277)
  Week 30; n=30,14: number analyzed (Participants) | 30 | 14
  Week 30; n=30,14 | -5.38 (95.013) | -4.66 (59.940)
  Week 36; n=16,6: number analyzed (Participants) | 16 | 6
  Week 36; n=16,6 | -1.55 (91.218) | 28.61 (86.861)

38. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage Changes From Baseline in Daily Average Number of Nocturia Episodes
Description: as for outcome 36
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: FAS3 Population. All the participants in this population were analyzed (56, 43 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percent change
  Week 0; n=54,38: number analyzed (Participants) | 54 | 38
  Week 0; n=54,38 | -10.30 (56.988) | -12.92 (66.778)
  Week 2; n=53,38: number analyzed (Participants) | 53 | 38
  Week 2; n=53,38 | -12.65 (56.372) | -17.41 (72.146)
  Week 6; n=51,37: number analyzed (Participants) | 51 | 37
  Week 6; n=51,37 | -10.34 (58.618) | -15.84 (67.482)
  Week 12; n=51,37: number analyzed (Participants) | 51 | 37
  Week 12; n=51,37 | -17.59 (58.516) | -23.85 (69.048)
  Week 18; n=21,26: number analyzed (Participants) | 21 | 26
  Week 18; n=21,26 | -2.77 (66.950) | -13.64 (71.573)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | 50.00 (70.711) | 16.73 (128.469)

39. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Severe Urgency Episodes
Description: The daily average number of urgency episodes categorized by each urgency intensity as no urgency, mild urgency, moderate urgency and severe urgency. Urgency episodes were calculated by a 4-point scale ranging from '0' (No urgency) to '3' (Severe urgency), as part of the bladder diary, during the 3-day diary collection period. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline in daily average number of severe urgency episodes was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.56 (2.702) | -1.72 (3.216)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -0.56 (2.737) | -1.92 (3.992)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.11 (2.624) | -1.98 (3.856)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -0.49 (3.141) | -2.02 (3.597)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -1.57 (4.441) | -1.69 (2.983)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -1.93 (4.636) | -1.59 (2.877)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -1.78 (5.426) | -1.53 (2.331)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -0.58 (3.646) | -1.46 (2.935)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -1.24 (4.600) | -1.52 (2.941)

40. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Severe Urgency Episodes
Description: as for outcome 39
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.00 (2.698) | -1.90 (3.799)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -2.11 (2.822) | -2.26 (4.424)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -1.89 (2.850) | -2.37 (3.952)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -1.69 (2.952) | -2.52 (4.031)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -1.58 (3.171) | -1.92 (3.794)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -1.78 (3.194) | -3.00 (4.603)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -1.56 (3.412) | -3.27 (4.823)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -2.03 (3.707) | -1.00 (3.502)

41. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Severe Urgency Episodes
Description: as for outcome 39
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -1.58 (2.357) | -3.05 (4.381)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -1.66 (2.658) | -3.52 (4.843)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -1.42 (2.245) | -3.41 (4.901)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -1.24 (2.350) | -3.24 (4.814)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -1.32 (2.466) | -3.28 (5.587)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -0.83 (1.179) | -1.92 (1.424)

42. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Daily Average Number of Severe or Moderate Urgency Episodes
Description: The daily average number of urgency episodes categorized by each urgency intensity as no urgency, mild urgency, moderate urgency and severe urgency. Urgency episodes were calculated by a 4-point scale ranging from '0' (No urgency), '1' (mild urgency), '2' (moderate urgency), '3' (Severe urgency), as part of the bladder diary, during the 3-day diary collection period. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day. Change from Baseline in daily average number of severe or moderate urgency episodes was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Episodes
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | -0.99 (3.097) | -2.28 (4.692)
  Week 6; n=124, 120: number analyzed (Participants) | 124 | 120
  Week 6; n=124, 120 | -1.17 (3.290) | -3.02 (4.376)
  Week 12; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12; n=122, 122 | -0.67 (3.330) | -2.89 (4.269)
  Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; n=23, 64 | -1.43 (3.441) | -3.16 (4.263)
  Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; n=17, 52 | -2.00 (3.629) | -3.51 (4.645)
  Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; n=14, 46 | -2.98 (3.037) | -3.18 (4.759)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -2.83 (4.707) | -3.16 (4.061)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -1.94 (4.685) | -3.21 (3.688)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -1.91 (3.944) | -2.58 (4.353)

43. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in Daily Average Number of Severe or Moderate Urgency Episodes
Description: as for outcome 42
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Episodes
  Week 0; n=108,88 | -0.40 (3.300) | -2.71 (3.874)
  Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; n=105,87 | -3.35 (3.819) | -3.39 (4.467)
  Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; n=106,84 | -3.19 (4.063) | -3.34 (3.890)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -3.10 (3.785) | -3.29 (3.663)
  Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; n=83,46 | -3.03 (3.626) | -2.76 (4.202)
  Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; n=45,21 | -3.33 (3.980) | -3.44 (3.015)
  Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; n=36,15 | -2.73 (5.063) | -3.62 (3.354)
  Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; n=20,6 | -4.12 (4.747) | -1.22 (4.698)

44. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in Daily Average Number of Severe or Moderate Urgency Episodes
Description: as for outcome 42
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Episodes
  Week 0; n=56,43 | -2.11 (3.132) | -3.39 (4.082)
  Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; n=55,43 | -2.47 (3.603) | -4.09 (4.104)
  Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; n=53,42 | -2.58 (2.819) | -4.18 (3.842)
  Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; n=53,41 | -2.23 (2.734) | -3.50 (3.936)
  Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; n=22,29 | -1.89 (3.155) | -2.98 (4.134)
  Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; n=2,4 | -3.33 (0.000) | -3.33 (4.815)

45. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Maximum Urgency Intensity
Description: The daily average number of urgency episodes categorized by each urgency intensity as no urgency (None), mild urgency, moderate urgency and severe urgency. Urgency episodes were calculated by a 4-point scale ranging from '0' (No urgency) to '3' (Severe urgency), as part of the bladder diary, during the 3-day diary collection period. "Maximum" was defined as the maximum urgency intensity within 3-day period (but only for valid diary day) in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day.
Time Frame: as for outcome 3
Population: FAS1 Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  None; Baseline (Pre-dose, Day 1); n=124, 124 | 0 | 0
  Mild; Baseline (Pre-dose, Day 1); n=124, 124 | 1 | 3
  Moderate; Baseline (Pre-dose, Day 1); n=124, 124 | 24 | 16
  Severe; Baseline (Pre-dose, Day 1); n=124, 124 | 99 | 105
  None; Week 2; n=124, 124 | 1 | 6
  Mild; Week 2; n=124, 124 | 11 | 21
  Moderate; Week 2; n=124, 124 | 25 | 36
  Severe; Week 2; n=124, 124 | 87 | 61
  None; Week 6; n=124, 124 | 1 | 15
  Mild; Week 6; n=124, 124 | 14 | 20
  Moderate; Week 6; n=124, 124 | 23 | 32
  Severe; Week 6; n=124, 124 | 86 | 57
  None; Week 12; n=124, 124 | 3 | 8
  Mild; Week 12; n=124, 124 | 9 | 16
  Moderate; Week 12; n=124, 124 | 22 | 37
  Severe; Week 12; n=124, 124 | 90 | 63
  None; Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  None; Week 18; n=23, 64 | 1 | 12
  Mild; Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Mild; Week 18; n=23, 64 | 3 | 11
  Moderate; Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Moderate; Week 18; n=23, 64 | 7 | 19
  Severe; Week 18; n=23, 64: number analyzed (Participants) | 23 | 64
  Severe; Week 18; n=23, 64 | 12 | 22
  None; Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  None; Week 24; n=17, 52 | 1 | 10
  Mild; Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Mild; Week 24; n=17, 52 | 1 | 10
  Moderate; Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Moderate; Week 24; n=17, 52 | 7 | 12
  Severe; Week 24; n=17, 52: number analyzed (Participants) | 17 | 52
  Severe; Week 24; n=17, 52 | 8 | 20
  None; Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  None; Week 30; n=14, 46 | 1 | 9
  Mild; Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Mild; Week 30; n=14, 46 | 3 | 8
  Moderate; Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Moderate; Week 30; n=14, 46 | 4 | 13
  Severe; Week 30; n=14, 46: number analyzed (Participants) | 14 | 46
  Severe; Week 30; n=14, 46 | 6 | 16
  None; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  None; Week 36; n=12, 32 | 1 | 8
  Mild; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Mild; Week 36; n=12, 32 | 2 | 4
  Moderate; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Moderate; Week 36; n=12, 32 | 5 | 9
  Severe; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Severe; Week 36; n=12, 32 | 4 | 11
  None; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  None; Week 42; n=11, 27 | 1 | 6
  Mild; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Mild; Week 42; n=11, 27 | 2 | 4
  Moderate; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Moderate; Week 42; n=11, 27 | 5 | 7
  Severe; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Severe; Week 42; n=11, 27 | 3 | 10
  None; Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  None; Week 48; n=11, 27 | 1 | 6
  Mild; Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Mild; Week 48; n=11, 27 | 1 | 3
  Moderate; Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Moderate; Week 48; n=11, 27 | 6 | 9
  Severe; Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Severe; Week 48; n=11, 27 | 3 | 9

46. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Number of Participants With Maximum Urgency Intensity
Description: The daily average number of urgency episodes categorized by each urgency intensity as no urgency (None), mild urgency, moderate urgency and severe urgency. Urgency episodes were calculated by a 4-point scale ranging from '0' (No urgency) to '3' (Severe urgency), as part of the bladder diary, during the 3-day diary collection period. "Maximum" was defined as the maximum urgency intensity within 3-day period (but only for valid diary day) in the visit.
Time Frame: Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30 and Week 36 in Treatment Cycle 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Participants
  None; Week 0; n=108,88 | 0 | 0
  Mild; Week 0; n=108,88 | 6 | 10
  Moderate; Week 0; n=108,88 | 20 | 24
  Severe; Week 0; n=108,88 | 82 | 54
  None; Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  None; Week 2; n=105,87 | 12 | 8
  Mild; Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Mild; Week 2; n=105,87 | 21 | 17
  Moderate; Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Moderate; Week 2; n=105,87 | 35 | 24
  Severe; Week 2; n=105,87: number analyzed (Participants) | 105 | 87
  Severe; Week 2; n=105,87 | 37 | 38
  None; Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  None; Week 6; n=106,84 | 13 | 9
  Mild; Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Mild; Week 6; n=106,84 | 27 | 12
  Moderate; Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Moderate; Week 6; n=106,84 | 25 | 27
  Severe; Week 6; n=106,84: number analyzed (Participants) | 106 | 84
  Severe; Week 6; n=106,84 | 41 | 36
  None; Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  None; Week 12; n=106,85 | 13 | 5
  Mild; Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Mild; Week 12; n=106,85 | 23 | 11
  Moderate; Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Moderate; Week 12; n=106,85 | 28 | 25
  Severe; Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Severe; Week 12; n=106,85 | 42 | 44
  None; Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  None; Week 18; n=83,46 | 11 | 5
  Mild; Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Mild; Week 18; n=83,46 | 16 | 8
  Moderate; Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Moderate; Week 18; n=83,46 | 21 | 10
  Severe; Week 18; n=83,46: number analyzed (Participants) | 83 | 46
  Severe; Week 18; n=83,46 | 35 | 23
  None; Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  None; Week 24; n=45,21 | 13 | 5
  Mild; Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Mild; Week 24; n=45,21 | 8 | 1
  Moderate; Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Moderate; Week 24; n=45,21 | 15 | 6
  Severe; Week 24; n=45,21: number analyzed (Participants) | 45 | 21
  Severe; Week 24; n=45,21 | 9 | 9
  None; Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  None; Week 30; n=36,15 | 9 | 3
  Mild; Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Mild; Week 30; n=36,15 | 6 | 3
  Moderate; Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Moderate; Week 30; n=36,15 | 10 | 1
  Severe; Week 30; n=36,15: number analyzed (Participants) | 36 | 15
  Severe; Week 30; n=36,15 | 11 | 8
  None; Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  None; Week 36; n=20,6 | 7 | 1
  Mild; Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Mild; Week 36; n=20,6 | 4 | 1
  Moderate; Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Moderate; Week 36; n=20,6 | 2 | 1
  Severe; Week 36; n=20,6: number analyzed (Participants) | 20 | 6
  Severe; Week 36; n=20,6 | 7 | 3

47. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Number of Participants With Maximum Urgency Intensity
Description: as for outcome 46
Time Frame: Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Participants
  None; Week 0; n=56,43 | 0 | 0
  Mild; Week 0; n=56,43 | 6 | 2
  Moderate; Week 0; n=56,43 | 14 | 16
  Severe; Week 0; n=56,43 | 36 | 25
  None; Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  None; Week 2; n=55,43 | 2 | 2
  Mild; Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Mild; Week 2; n=55,43 | 6 | 5
  Moderate; Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Moderate; Week 2; n=55,43 | 15 | 19
  Severe; Week 2; n=55,43: number analyzed (Participants) | 55 | 43
  Severe; Week 2; n=55,43 | 32 | 17
  None; Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  None; Week 6; n=53,42 | 3 | 3
  Mild; Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Mild; Week 6; n=53,42 | 10 | 5
  Moderate; Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Moderate; Week 6; n=53,42 | 12 | 15
  Severe; Week 6; n=53,42: number analyzed (Participants) | 53 | 42
  Severe; Week 6; n=53,42 | 28 | 19
  None; Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  None; Week 12; n=53,41 | 3 | 3
  Mild; Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Mild; Week 12; n=53,41 | 8 | 5
  Moderate; Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Moderate; Week 12; n=53,41 | 9 | 14
  Severe; Week 12; n=53,41: number analyzed (Participants) | 53 | 41
  Severe; Week 12; n=53,41 | 33 | 19
  None; Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  None; Week 18; n=22,29 | 2 | 1
  Mild; Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Mild; Week 18; n=22,29 | 3 | 4
  Moderate; Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Moderate; Week 18; n=22,29 | 5 | 9
  Severe; Week 18; n=22,29: number analyzed (Participants) | 22 | 29
  Severe; Week 18; n=22,29 | 12 | 15
  None; Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  None; Week 24; n=2,4 | 0 | 0
  Mild; Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Mild; Week 24; n=2,4 | 0 | 0
  Moderate; Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Moderate; Week 24; n=2,4 | 0 | 2
  Severe; Week 24; n=2,4: number analyzed (Participants) | 2 | 4
  Severe; Week 24; n=2,4 | 2 | 2

48. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Improvement and Worsening in Maximum Urgency Intensity From Baseline
Description: Urgency intensity was determined using a 4-point scale ranging from 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe) as part of the bladder diary, during the 3-day diary collection period. "Maximum" was defined as the maximum urgency intensity within 3-day period (but only for valid diary day) in the visit. Results have been presented for improvement (3 point, 2 point, 1 point improvement and no change) as well as for worsening (1 point, 2 point, 3 point worsening) of urgency intensity. Maximum possible scale range is 0 to 3. 3 point improvement means change in intensity from severe to none. 3 point worsening means change in intensity from none to severe. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day.
Time Frame: as for outcome 3
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Week 2; 3 point improvement; n=124, 124 | 0 | 5
  Week 2; 2 point improvement; n=124, 124 | 5 | 13
  Week 2; 1 point improvement; n=124, 124 | 19 | 35
  Week 2; No change; n=124, 124 | 95 | 69
  Week 6; 3 point improvement; n=124, 124 | 0 | 12
  Week 6; 2 point improvement; n=124, 124 | 5 | 15
  Week 6; 1 point improvement; n=124, 124 | 24 | 31
  Week 6; No change; n=124, 124 | 89 | 64
  Week 12; 3 point improvement; n=124, 124 | 3 | 5
  Week 12; 2 point improvement; n=124, 124 | 2 | 12
  Week 12; 1 point improvement; n=124, 124 | 20 | 36
  Week 12; No change; n=124, 124 | 89 | 67
  Week 18; 3 point improvement; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 3 point improvement; n=23, 64 | 1 | 8
  Week 18; 2 point improvement; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 2 point improvement; n=23, 64 | 2 | 9
  Week 18; 1 point improvement; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 1 point improvement; n=23, 64 | 4 | 25
  Week 18; No change; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; No change; n=23, 64 | 15 | 20
  Week 24; 3 point improvement; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 3 point improvement; n=17, 52 | 1 | 8
  Week 24; 2 point improvement; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 2 point improvement; n=17, 52 | 1 | 8
  Week 24; 1 point improvement; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 1 point improvement; n=17, 52 | 4 | 13
  Week 24; No change; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; No change; n=17, 52 | 11 | 23
  Week 30; 3 point improvement; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 3 point improvement; n=14, 46 | 1 | 7
  Week 30; 2 point improvement; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 2 point improvement; n=14, 46 | 3 | 8
  Week 30; 1 point improvement; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 1 point improvement; n=14, 46 | 2 | 12
  Week 30; No change; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; No change; n=14, 46 | 8 | 17
  Week 36; 3 point improvement; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 3 point improvement; n=12, 32 | 1 | 5
  Week 36; 2 point improvement; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 2 point improvement; n=12, 32 | 2 | 5
  Week 36; 1 point improvement; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 1 point improvement; n=12, 32 | 3 | 9
  Week 36; No change; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; No change; n=12, 32 | 6 | 12
  Week 42; 3 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 3 point improvement; n=11, 27 | 1 | 2
  Week 42; 2 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 2 point improvement; n=11, 27 | 2 | 6
  Week 42; 1 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 1 point improvement; n=11, 27 | 3 | 9
  Week 42; No change; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; No change; n=11, 27 | 5 | 9
  Week 48; 3 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 3 point improvement; n=11, 27 | 1 | 3
  Week 48; 2 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 2 point improvement; n=11, 27 | 1 | 4
  Week 48; 1 point improvement; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 1 point improvement; n=11, 27 | 4 | 10
  Week 48; No change; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; No change; n=11, 27 | 5 | 9
  Week 2; 1 point worsening; n=124, 124 | 5 | 2
  Week 2; 2 point worsening; n=124, 124 | 0 | 0
  Week 2; 3 point worsening; n=124, 124 | 0 | 0
  Week 6; 1 point worsening; n=124, 124 | 6 | 2
  Week 6;2 point worsening; n=124, 124 | 0 | 0
  Week 6; 3 point worsening; n=124, 124 | 0 | 0
  Week 12; 1 point worsening; n=124, 124 | 10 | 4
  Week 12; 2 point worsening; n=124, 124 | 0 | 0
  Week 12; 3 point worsening; n=124, 124 | 0 | 0
  Week 18; 1 point worsening; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 1 point worsening; n=23, 64 | 1 | 2
  Week 18; 2 point worsening; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 2 point worsening; n=23, 64 | 0 | 0
  Week 18; 3 point worsening; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 3 point worsening; n=23, 64 | 0 | 0
  Week 24; 1 point worsening; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 1 point worsening; n=17, 52 | 0 | 0
  Week 24; 2 point worsening; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 2 point worsening; n=17, 52 | 0 | 0
  Week 24; 3 point worsening; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 3 point worsening; n=17, 52 | 0 | 0
  Week 30; 1 point worsening; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 1 point worsening; n=14, 46 | 0 | 2
  Week 30; 2 point worsening; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 2 point worsening; n=14, 46 | 0 | 0
  Week 30; 3 point worsening; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 3 point worsening; n=14, 46 | 0 | 0
  Week 36; 1 point worsening; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 1 point worsening; n=12, 32 | 0 | 1
  Week 36; 2 point worsening; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 2 point worsening; n=12, 32 | 0 | 0
  Week 36; 3 point worsening; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 3 point worsening; n=12, 32 | 0 | 0
  Week 42; 1 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 1 point worsening; n=11, 27 | 0 | 1
  Week 42; 2 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 2 point worsening; n=11, 27 | 0 | 0
  Week 42; 3 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 3 point worsening; n=11, 27 | 0 | 0
  Week 48; 1 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 1 point worsening; n=11, 27 | 0 | 1
  Week 48; 2 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 2 point worsening; n=11, 27 | 0 | 0
  Week 48; 3 point worsening; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 3 point worsening; n=11, 27 | 0 | 0

49. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Number of Participants With Improvement and Worsening in Maximum Urgency Intensity From Baseline
Description: as for outcome 48
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Participants
  Week 0; 3 point improvement; n=108,88 | 0 | 0
  Week 0; 2 point improvement; n=108,88 | 1 | 6
  Week 0; 1 point improvement; n=108,88 | 16 | 24
  Week 0; No change; n=108,88 | 83 | 54
  Week 2; 3 point improvement; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; 3 point improvement; n=105,87 | 10 | 5
  Week 2; 2 point improvement; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; 2 point improvement; n=105,87 | 14 | 14
  Week 2; 1 point improvement; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; 1 point improvement; n=105,87 | 37 | 27
  Week 2; No change; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; No change; n=105,87 | 41 | 41
  Week 6; 3 point improvement; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; 3 point improvement; n=106,84 | 10 | 7
  Week 6; 2 point improvement; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; 2 point improvement; n=106,84 | 20 | 8
  Week 6; 1 point improvement; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; 1 point improvement; n=106,84 | 29 | 32
  Week 6; No change; n=106,84: number analyzed (Participants) | 106 | 84
  Week 6; No change; n=106,84 | 44 | 34
  Week 12; 3 point improvement; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; 3 point improvement; n=106,85 | 9 | 4
  Week 12; 2 point improvement; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; 2 point improvement; n=106,85 | 17 | 7
  Week 12; 1 point improvement; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; 1 point improvement; n=106,85 | 31 | 27
  Week 12; No change;n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; No change;n=106,85 | 48 | 44
  Week 18; 3 point improvement; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; 3 point improvement; n=83,46 | 6 | 4
  Week 18; 2 point improvement; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; 2 point improvement; n=83,46 | 14 | 6
  Week 18; 1 point improvement; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; 1 point improvement; n=83,46 | 23 | 12
  Week 18; No change; n=83,46: number analyzed (Participants) | 83 | 46
  Week 18; No change; n=83,46 | 37 | 22
  Week 24; 3 point improvement; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; 3 point improvement; n=45,21 | 7 | 2
  Week 24; 2 point improvement; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; 2 point improvement; n=45,21 | 11 | 4
  Week 24; 1 point improvement; n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; 1 point improvement; n=45,21 | 12 | 6
  Week 24; No change;n=45,21: number analyzed (Participants) | 45 | 21
  Week 24; No change;n=45,21 | 15 | 9
  Week 30; 3 point improvement; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; 3 point improvement; n=36,15 | 7 | 2
  Week 30; 2 point improvement; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; 2 point improvement; n=36,15 | 5 | 3
  Week 30; 1 point improvement; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; 1 point improvement; n=36,15 | 10 | 2
  Week 30; No change; n=36,15: number analyzed (Participants) | 36 | 15
  Week 30; No change; n=36,15 | 13 | 8
  Week 36; 3 point improvement; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; 3 point improvement; n=20,6 | 5 | 1
  Week 36; 2 point improvement; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; 2 point improvement; n=20,6 | 6 | 1
  Week 36; 1 point improvement; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; 1 point improvement; n=20,6 | 1 | 0
  Week 36; No change; n=20,6: number analyzed (Participants) | 20 | 6
  Week 36; No change; n=20,6 | 8 | 4
  Week 0; 1 point worsening; n=108,88 | 8 | 4
  Week 0; 2 point worsening; n=108,88 | 0 | 0
  Week 0; 3 point worsening; n=108,88 | 0 | 0
  Week 2; 1 point worsening; n=105,87: number analyzed (Participants) | 105 | 87
  Week 2; 1 point worsening; n=105,87 | 3 | 0
  Week 2; 2 point worsening; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; 2 point worsening; n=105, 87 | 0 | 0
  Week 2; 3 point worsening; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; 3 point worsening; n=105, 87 | 0 | 0
  Week 6; 1 point worsening; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; 1 point worsening; n=106, 84 | 3 | 3
  Week 6;2 point worsening; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6;2 point worsening; n=106, 84 | 0 | 0
  Week 6; 3 point worsening; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; 3 point worsening; n=106, 84 | 0 | 0
  Week 12; 1 point worsening; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; 1 point worsening; n=106, 85 | 1 | 3
  Week 12; 2 point worsening; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; 2 point worsening; n=106, 85 | 0 | 0
  Week 12; 3 point worsening; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; 3 point worsening; n=106, 85 | 0 | 0
  Week 18; 1 point worsening; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; 1 point worsening; n=83, 46 | 3 | 2
  Week 18; 2 point worsening; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; 2 point worsening; n=83, 46 | 0 | 0
  Week 18; 3 point worsening; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; 3 point worsening; n=83, 46 | 0 | 0
  Week 24; 1 point worsening; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; 1 point worsening; n=45, 21 | 0 | 0
  Week 24; 2 point worsening; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; 2 point worsening; n=45, 21 | 0 | 0
  Week 24; 3 point worsening; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; 3 point worsening; n=45, 21 | 0 | 0
  Week 30; 1 point worsening; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; 1 point worsening; n=36, 15 | 1 | 0
  Week 30; 2 point worsening; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; 2 point worsening; n=36, 15 | 0 | 0
  Week 30; 3 point worsening; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; 3 point worsening; n=36, 15 | 0 | 0
  Week 36; 1 point worsening; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; 1 point worsening; n=20, 6 | 0 | 0
  Week 36; 2 point worsening; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; 2 point worsening; n=20, 6 | 0 | 0
  Week 36; 3 point worsening; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; 3 point worsening; n=20, 6 | 0 | 0

50. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Number of Participants With Improvement and Worsening in Maximum Urgency Intensity From Baseline
Description: as for outcome 48
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Participants
  Week 0; 3 point improvement; n=56,43 | 0 | 0
  Week 0; 2 point improvement; n=56,43 | 3 | 1
  Week 0; 1 point improvement; n=56,43 | 13 | 14
  Week 0; No change; n=56,43 | 39 | 26
  Week 2; 3 point improvement; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 3 point improvement; n=55,43 | 2 | 1
  Week 2; 2 point improvement; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 2 point improvement; n=55,43 | 3 | 5
  Week 2; 1 point improvement; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 1 point improvement; n=55,43 | 13 | 19
  Week 2; No change; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; No change; n=55,43 | 37 | 15
  Week 6; 3 point improvement; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; 3 point improvement; n=53,42 | 1 | 3
  Week 6; 2 point improvement; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; 2 point improvement; n=53,42 | 7 | 4
  Week 6; 1 point improvement; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; 1 point improvement; n=53,42 | 16 | 12
  Week 6; No change; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; No change; n=53,42 | 29 | 22
  Week 12; 3 point improvement; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; 3 point improvement; n=53,41 | 2 | 2
  Week 12; 2 point improvement; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; 2 point improvement; n=53,41 | 5 | 5
  Week 12; 1 point improvement; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; 1 point improvement; n=53,41 | 10 | 13
  Week 12; No change;n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; No change;n=53,41 | 36 | 20
  Week 18; 3 point improvement; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; 3 point improvement; n=22,29 | 2 | 1
  Week 18; 2 point improvement; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; 2 point improvement; n=22,29 | 1 | 3
  Week 18; 1 point improvement; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; 1 point improvement; n=22,29 | 4 | 7
  Week 18; No change; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; No change; n=22,29 | 15 | 18
  Week 24; 3 point improvement; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; 3 point improvement; n=2,4 | 0 | 0
  Week 24; 2 point improvement; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; 2 point improvement; n=2,4 | 0 | 0
  Week 24; 1 point improvement; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; 1 point improvement; n=2,4 | 0 | 2
  Week 24; No change;n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; No change;n=2,4 | 2 | 2
  Week 0; 1 point worsening; n=56,43 | 1 | 2
  Week 0; 2 point worsening; n=56,43 | 0 | 0
  Week 0; 3 point worsening; n=56,43 | 0 | 0
  Week 2; 1 point worsening; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 1 point worsening; n=55,43 | 0 | 3
  Week 2; 2 point worsening; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 2 point worsening; n=55,43 | 0 | 0
  Week 2; 3 point worsening; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 3 point worsening; n=55,43 | 0 | 0
  Week 6; 1 point worsening; n=53, 42: number analyzed (Participants) | 53 | 42
  Week 6; 1 point worsening; n=53, 42 | 0 | 1
  Week 6;2 point worsening; n=53, 42: number analyzed (Participants) | 53 | 42
  Week 6;2 point worsening; n=53, 42 | 0 | 0
  Week 6; 3 point worsening; n=53, 42: number analyzed (Participants) | 53 | 42
  Week 6; 3 point worsening; n=53, 42 | 0 | 0
  Week 12; 1 point worsening; n=53, 41: number analyzed (Participants) | 53 | 41
  Week 12; 1 point worsening; n=53, 41 | 0 | 1
  Week 12; 2 point worsening; n=53, 41: number analyzed (Participants) | 53 | 41
  Week 12; 2 point worsening; n=53, 41 | 0 | 0
  Week 12; 3 point worsening; n=53, 41: number analyzed (Participants) | 53 | 41
  Week 12; 3 point worsening; n=53, 41 | 0 | 0
  Week 18; 1 point worsening; n=22, 29: number analyzed (Participants) | 22 | 29
  Week 18; 1 point worsening; n=22, 29 | 0 | 0
  Week 18; 2 point worsening; n=22, 29: number analyzed (Participants) | 22 | 29
  Week 18; 2 point worsening; n=22, 29 | 0 | 0
  Week 18; 3 point worsening; n=22, 29: number analyzed (Participants) | 22 | 29
  Week 18; 3 point worsening; n=22, 29 | 0 | 0
  Week 24; 1 point worsening; n=2, 4: number analyzed (Participants) | 2 | 4
  Week 24; 1 point worsening; n=2, 4 | 0 | 0
  Week 24; 2 point worsening; n=2, 4: number analyzed (Participants) | 2 | 4
  Week 24; 2 point worsening; n=2, 4 | 0 | 0
  Week 24; 3 point worsening; n=2, 4: number analyzed (Participants) | 2 | 4
  Week 24; 3 point worsening; n=2, 4 | 0 | 0

51. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage of Participants Attaining 100 Percent (%), >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1)", excluding the day of visit (this period was called the '3-day diary collection period'). The daily average of the number of incontinence episodes were calculated using formula; number of "Yes" response to the diary question of "Did you have accidental urinary leakage?" divided by number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day.
Time Frame: as for outcome 3
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percentage of participants
  Week 2; 100 %; n=124, 124 | 3 | 18
  Week 2; >=75%; n=124, 124 | 9 | 40
  Week 2; >=50%; n=124, 124 | 23 | 55
  Week 6; 100 %; n=124, 124 | 3 | 27
  Week 6; >=75%; n=124, 124 | 8 | 41
  Week 6; >=50%; n=124, 124 | 27 | 60
  Week 12; 100 %; n=124, 124 | 3 | 19
  Week 12; >=75%; n=124, 124 | 14 | 40
  Week 12; >=50%; n=124, 124 | 24 | 58
  Week 18; 100 %; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 100 %; n=23, 64 | 13 | 33
  Week 18; >=75%; n= 23, 64: number analyzed (Participants) | 23 | 64
  Week 18; >=75%; n= 23, 64 | 35 | 56
  Week 18; >=50%; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; >=50%; n=23, 64 | 52 | 66
  Week 24; 100 %; n= 17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 100 %; n= 17, 52 | 24 | 38
  Week 24; >=75%; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; >=75%; n=17, 52 | 53 | 63
  Week 24; >=50%; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; >=50%; n=17, 52 | 71 | 77
  Week 30; 100 %; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 100 %; n=14, 46 | 36 | 28
  Week 30; >=75%; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; >=75%; n=14, 46 | 57 | 52
  Week 30; >=50%; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; >=50%; n=14, 46 | 71 | 65
  Week 36; 100 %; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 100 %; n=12, 32 | 25 | 34
  Week 36; >=75%; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; >=75%; n=12, 32 | 58 | 50
  Week 36; >=50%; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; >=50%; n=12, 32 | 75 | 66
  Week 42; 100 %; n= 11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 100 %; n= 11, 27 | 18 | 33
  Week 42; >=75%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; >=75%; n=11, 27 | 55 | 56
  Week 42; >=50%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; >=50%; n=11, 27 | 64 | 70
  Week 48; 100 %; n= 11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 100 %; n= 11, 27 | 27 | 33
  Week 48; >=75%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; >=75%; n=11, 27 | 55 | 48
  Week 48; >=50%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; >=50%; n=11, 27 | 73 | 63

52. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: as for outcome 51
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percentage of participants
  Week 0; 100%; n=108,88 | 0 | 0
  Week 0; >=75%; n=108,88 | 6 | 17
  Week 0; >=50%; n=108,88 | 19 | 42
  Week 2; 100 %; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; 100 %; n=105, 87 | 30 | 20
  Week 2; >=75%; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; >=75%; n=105, 87 | 57 | 53
  Week 2; >=50%; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; >=50%; n=105, 87 | 81 | 71
  Week 6; 100 %; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; 100 %; n=106, 84 | 35 | 18
  Week 6; >=75%; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; >=75%; n=106, 84 | 58 | 57
  Week 6; >=50%; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; >=50%; n=106, 84 | 71 | 71
  Week 12; 100 %; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; 100 %; n=106, 85 | 27 | 19
  Week 12; >=75%; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; >=75%; n=106, 85 | 53 | 41
  Week 12; >=50%; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; >=50%; n=106, 85 | 74 | 64
  Week 18; 100 %; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; 100 %; n=83, 46 | 18 | 28
  Week 18; >=75%; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; >=75%; n=83, 46 | 43 | 43
  Week 18; >=50%; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; >=50%; n=83, 46 | 66 | 72
  Week 24; 100 %; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; 100 %; n=45, 21 | 40 | 38
  Week 24; >=75%; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; >=75%; n=45, 21 | 56 | 67
  Week 24; >=50%; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; >=50%; n=45, 21 | 71 | 86
  Week 30; 100 %; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; 100 %; n=36, 15 | 22 | 40
  Week 30; >=75%; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; >=75%; n=36, 15 | 53 | 47
  Week 30; >=50%; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; >=50%; n=36, 15 | 75 | 80
  Week 36; 100 %; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; 100 %; n=20, 6 | 45 | 33
  Week 36; >=75%; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; >=75%; n=20, 6 | 55 | 67
  Week 36; >=50%; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; >=50%; n=20, 6 | 75 | 67

53. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: as for outcome 51
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percentage of participants
  Week 0; 100%; n=56,43 | 0 | 0
  Week 0; >=75%; n=56,43 | 21 | 7
  Week 0; >=50%; n=56,43 | 50 | 40
  Week 2; 100 %; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 100 %; n=55,43 | 13 | 16
  Week 2; >=75%; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; >=75%; n=55,43 | 36 | 42
  Week 2; >=50%; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; >=50%; n=55,43 | 64 | 58
  Week 6; 100 %; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; 100 %; n=53,42 | 13 | 12
  Week 6; >=75%; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; >=75%; n=53,42 | 43 | 43
  Week 6; >=50%; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; >=50%; n=53,42 | 70 | 76
  Week 12; 100 %; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; 100 %; n=53,41 | 13 | 10
  Week 12; >=75%; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; >=75%; n=53,41 | 45 | 34
  Week 12; >=50%; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; >=50%; n=53,41 | 62 | 54
  Week 18; 100 %; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; 100 %; n=22,29 | 18 | 3
  Week 18; >=75%; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; >=75%; n=22,29 | 18 | 34
  Week 18; >=50%; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; >=50%; n=22,29 | 50 | 55
  Week 24; 100 %; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; 100 %; n=2,4 | 0 | 0
  Week 24; >=75%; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; >=75%; n=2,4 | 0 | 0
  Week 24; >=50%; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; >=50%; n=2,4 | 0 | 50

54. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Urgency Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1)", excluding the day of visit (this period was called the '3-day diary collection period'). The daily average number of urge incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage and sudden/ urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day.
Time Frame: as for outcome 3
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percentage of participants
  Week 2; 100 %; n=124, 124 | 3 | 19
  Week 2; >=75%; n=124, 124 | 10 | 44
  Week 2; >=50%; n=124, 124 | 25 | 56
  Week 6; 100 %; n=124, 124 | 4 | 30
  Week 6; >=75%; n=124, 124 | 9 | 44
  Week 6; >=50%; n=124, 124 | 27 | 61
  Week 12; 100 %; n=124, 124 | 5 | 21
  Week 12; >=75%; n=124, 124 | 13 | 42
  Week 12; >=50%; n=124, 124 | 26 | 58
  Week 18; 100 %; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; 100 %; n=23, 64 | 13 | 36
  Week 18; >=75%; n= 23, 64: number analyzed (Participants) | 23 | 64
  Week 18; >=75%; n= 23, 64 | 35 | 56
  Week 18; >=50%; n=23, 64: number analyzed (Participants) | 23 | 64
  Week 18; >=50%; n=23, 64 | 52 | 67
  Week 24; 100 %; n= 17, 52: number analyzed (Participants) | 17 | 52
  Week 24; 100 %; n= 17, 52 | 29 | 40
  Week 24; >=75%; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; >=75%; n=17, 52 | 53 | 67
  Week 24; >=50%; n=17, 52: number analyzed (Participants) | 17 | 52
  Week 24; >=50%; n=17, 52 | 76 | 81
  Week 30; 100 %; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; 100 %; n=14, 46 | 43 | 30
  Week 30; >=75%; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; >=75%; n=14, 46 | 64 | 54
  Week 30; >=50%; n=14, 46: number analyzed (Participants) | 14 | 46
  Week 30; >=50%; n=14, 46 | 71 | 70
  Week 36; 100 %; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; 100 %; n=12, 32 | 25 | 38
  Week 36; >=75%; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; >=75%; n=12, 32 | 58 | 53
  Week 36; >=50%; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; >=50%; n=12, 32 | 75 | 72
  Week 42; 100 %; n= 11, 27: number analyzed (Participants) | 11 | 27
  Week 42; 100 %; n= 11, 27 | 18 | 44
  Week 42; >=75%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; >=75%; n=11, 27 | 64 | 67
  Week 42; >=50%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; >=50%; n=11, 27 | 73 | 81
  Week 48; 100 %; n= 11, 27: number analyzed (Participants) | 11 | 27
  Week 48; 100 %; n= 11, 27 | 36 | 37
  Week 48; >=75%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; >=75%; n=11, 27 | 64 | 56
  Week 48; >=50%; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; >=50%; n=11, 27 | 82 | 78

55. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Urgency Incontinence Episodes
Description: as for outcome 54
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percentage of participants
  Week 0; 100%; n=108,88 | 0 | 0
  Week 0; >=75%; n=108,88 | 6 | 17
  Week 0; >=50%; n=108,88 | 19 | 42
  Week 2; 100 %; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; 100 %; n=105, 87 | 31 | 24
  Week 2; >=75%; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; >=75%; n=105, 87 | 57 | 56
  Week 2; >=50%; n=105, 87: number analyzed (Participants) | 105 | 87
  Week 2; >=50%; n=105, 87 | 80 | 72
  Week 6; 100 %; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; 100 %; n=106, 84 | 35 | 20
  Week 6; >=75%; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; >=75%; n=106, 84 | 59 | 57
  Week 6; >=50%; n=106, 84: number analyzed (Participants) | 106 | 84
  Week 6; >=50%; n=106, 84 | 71 | 71
  Week 12; 100 %; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; 100 %; n=106, 85 | 28 | 19
  Week 12; >=75%; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; >=75%; n=106, 85 | 55 | 42
  Week 12; >=50%; n=106, 85: number analyzed (Participants) | 106 | 85
  Week 12; >=50%; n=106, 85 | 73 | 64
  Week 18; 100 %; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; 100 %; n=83, 46 | 18 | 28
  Week 18; >=75%; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; >=75%; n=83, 46 | 45 | 43
  Week 18; >=50%; n=83, 46: number analyzed (Participants) | 83 | 46
  Week 18; >=50%; n=83, 46 | 65 | 74
  Week 24; 100 %; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; 100 %; n=45, 21 | 42 | 38
  Week 24; >=75%; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; >=75%; n=45, 21 | 56 | 67
  Week 24; >=50%; n=45, 21: number analyzed (Participants) | 45 | 21
  Week 24; >=50%; n=45, 21 | 73 | 86
  Week 30; 100 %; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; 100 %; n=36, 15 | 31 | 40
  Week 30; >=75%; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; >=75%; n=36, 15 | 61 | 47
  Week 30; >=50%; n=36, 15: number analyzed (Participants) | 36 | 15
  Week 30; >=50%; n=36, 15 | 75 | 80
  Week 36; 100 %; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; 100 %; n=20, 6 | 50 | 33
  Week 36; >=75%; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; >=75%; n=20, 6 | 60 | 67
  Week 36; >=50%; n=20, 6: number analyzed (Participants) | 20 | 6
  Week 36; >=50%; n=20, 6 | 75 | 67

56. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Urgency Incontinence Episodes
Description: Participants were instructed to enter data in a bladder diary over 3 consecutive days within a week prior to each scheduled visit (or within 28 days prior to Day 1)", excluding the day of visit (this period was called the '3-day diary collection period'). The daily average number of urge incontinence episodes were calculated from bladder diary data recorded by the participants during the 3-day diary collection period, by dividing the number of 'Yes' response to the diary question of accidental urinary leakage and sudden/urgent need to urinate with the number of valid diary days in the visit. Baseline is the latest pre-dose 3-day diary assessment which has at least one valid diary day.
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percentage of participants
  Week 0; 100%; n=56,43 | 0 | 0
  Week 0; >=75%; n=56,43 | 21 | 7
  Week 0; >=50%; n=56,43 | 48 | 40
  Week 2; 100 %; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; 100 %; n=55,43 | 16 | 19
  Week 2; >=75%; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; >=75%; n=55,43 | 35 | 42
  Week 2; >=50%; n=55,43: number analyzed (Participants) | 55 | 43
  Week 2; >=50%; n=55,43 | 67 | 60
  Week 6; 100 %; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; 100 %; n=53,42 | 15 | 14
  Week 6; >=75%; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; >=75%; n=53,42 | 47 | 43
  Week 6; >=50%; n=53,42: number analyzed (Participants) | 53 | 42
  Week 6; >=50%; n=53,42 | 68 | 69
  Week 12; 100 %; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; 100 %; n=53,41 | 15 | 12
  Week 12; >=75%; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; >=75%; n=53,41 | 47 | 37
  Week 12; >=50%; n=53,41: number analyzed (Participants) | 53 | 41
  Week 12; >=50%; n=53,41 | 64 | 59
  Week 18; 100 %; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; 100 %; n=22,29 | 18 | 3
  Week 18; >=75%; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; >=75%; n=22,29 | 23 | 38
  Week 18; >=50%; n=22,29: number analyzed (Participants) | 22 | 29
  Week 18; >=50%; n=22,29 | 55 | 59
  Week 24; 100 %; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; 100 %; n=2,4 | 0 | 0
  Week 24; >=75%; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; >=75%; n=2,4 | 0 | 0
  Week 24; >=50%; n=2,4: number analyzed (Participants) | 2 | 4
  Week 24; >=50%; n=2,4 | 0 | 50

57. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Time to Qualification for Retreatment
Description: Participants were considered for re-treatment beginning at the Week 12 visit following the initial treatment or the Week 12 visit following any re-treatment. Qualification criteria was; participants must have initiated request for re-treatment, participants experienced >=2 episodes of urinary urgency incontinence, with no more than one urgency incontinence-free day, post-void residual (PVR) urine volume must have been <200 milliliter; investigator deemed re-treatment appropriate. Time to the participant's first qualification for 2nd treatment from the day of 1st treatment was calculated as the earliest date when participants fulfilled the qualification for retreatment criteria minus the day of first treatment plus 1.
Time Frame: Up to 36 weeks in Treatment Cycle 1
Population: FAS1 Population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Days | 85.0 [84.0 to 85.0] | 127.0 [91.0 to 175.0]
Statistical Analysis 1: Comparison: Treatment Cycle 1: Placebo vs Treatment Cycle 1: GSK1358820 100 U; Test type: Other; p < 0.001, Log Rank — P-value is from log-rank test stratified by Baseline urinary urgency incontinence episodes over 3 day diary (<=9 versus >=10); Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.34 to 0.60] — Hazard ratio and 95% Confidence Interval (CI) are estimated using the Cox proportional hazard model with treatment and Baseline urinary urgency incontinence episodes over 3 day diary (<=9 versus >=10) as fixed effect

58. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Time to Request for Retreatment
Description: The time taken by the participants to request re-treatment was reported. Time to the participant's first request for 2nd treatment from the day of 1st treatment was calculated as the earliest date when participants requested retreatment minus the day of first treatment plus 1.
Time Frame: Up to 36 weeks in Treatment Cycle 1
Population: FAS1 Population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Days | 85.0 [84.0 to 85.0] | 92.0 [85.0 to 128.0]
Statistical Analysis 1: Comparison: Treatment Cycle 1: Placebo vs Treatment Cycle 1: GSK1358820 100 U; Test type: Other; p < 0.001, Log Rank — [p-value comment as in outcome 57, analysis 1]; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.66] — Hazard ratio and 95% CI are estimated using the Cox proportional hazard model with treatment and Baseline urinary urgency incontinence episodes over 3 day diary (<=9 versus >=10) as fixed effect

59. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in King's Health Questionnaire (KHQ) Domain Scores
Description: KHQ is a 21 item questionnaire, consisting of 9 domains: General health (GH) (1[Very good] to 5[Very poor]), Incontinence impact (Int Imp) (1[Not at all] to 4[A lot]), Role Limitations (RL) (1[Not at all] to 4[A lot]), Physical limitations (PL) (1[Not at all] to 4[A lot]), Social limitations (SL) (0[not applicable] to 4[A lot]), Personal relationships (PR) (0[Not applicable] to 4[A lot]), Emotions (1[Not at all] to 4[Very much]), Sleep/ energy (S/ E) (1[Never] to 4[All the time]) and Severity/Coping (S/ C) (1[Never] to 4[All the time]). Domain score for GH was calculated as score of one item minus 1/4x100; Int Imp: score of one item minus 1/3x100; RL, PL, PR, S/ E: summed scores of 2 items minus 2/6x100; SL, Emotions: summed scores of 3 items minus 3/9x100; S/ C: summed scores of 5 items minus 5/15x100. Baseline is the latest pre-dose assessment with a non-missing value,including those from unscheduled visits. Change from Baseline was any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Scores on a scale
  General Health Perception; Week 12;n=122, 123: number analyzed (Participants) | 122 | 123
  General Health Perception; Week 12;n=122, 123 | 4.9 (26.43) | -1.8 (24.41)
  General Health Perception; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  General Health Perception; Week 24;n=17, 54 | -10.3 (19.88) | -2.8 (17.95)
  General Health Perception; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  General Health Perception; Week 36;n=12, 32 | -10.4 (19.82) | -3.9 (18.08)
  General Health Perception; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  General Health Perception; Week 48;n=11, 27 | -6.8 (11.68) | 0.0 (19.61)
  Incontinence Impact; Week 12;n=122, 123: number analyzed (Participants) | 122 | 123
  Incontinence Impact; Week 12;n=122, 123 | -6.56 (27.320) | -23.04 (36.497)
  Incontinence Impact; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Incontinence Impact; Week 24;n=17, 54 | -25.49 (25.082) | -36.42 (32.550)
  Incontinence Impact; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Incontinence Impact; Week 36;n=12, 32 | -30.56 (17.164) | -43.75 (24.593)
  Incontinence Impact; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Incontinence Impact; Week 48;n=11, 27 | -27.27 (25.025) | -33.33 (24.460)
  Role Limitations; Week 12;n= 121, 123: number analyzed (Participants) | 121 | 123
  Role Limitations; Week 12;n= 121, 123 | -3.03 (24.814) | -18.56 (34.290)
  Role Limitations; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Role Limitations; Week 24;n=17, 54 | -8.82 (26.430) | -30.25 (32.710)
  Role Limitations; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Role Limitations; Week 36;n=12, 32 | -18.06 (25.084) | -26.04 (33.317)
  Role Limitations; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Role Limitations; Week 48;n=11, 27 | -15.15 (36.098) | -22.84 (33.059)
  Physical Limitations; Week 12;n=121, 123: number analyzed (Participants) | 121 | 123
  Physical Limitations; Week 12;n=121, 123 | -3.31 (26.581) | -15.18 (35.388)
  Physical Limitations; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Physical Limitations; Week 24;n=17, 54 | -13.73 (26.507) | -27.47 (33.515)
  Physical Limitations; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Physical Limitations; Week 36;n=12, 32 | -16.67 (29.302) | -24.48 (29.930)
  Physical Limitations; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Physical Limitations; Week 48;n=11, 27 | -16.67 (27.889) | -17.28 (32.186)
  Social Limitations; Week 12;n=121, 123: number analyzed (Participants) | 121 | 123
  Social Limitations; Week 12;n=121, 123 | -0.78 (25.952) | -11.92 (30.326)
  Social Limitations; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Social Limitations; Week 24;n=17, 54 | -12.75 (28.175) | -21.60 (34.019)
  Social Limitations; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Social Limitations; Week 36;n=12, 32 | -25.93 (30.089) | -18.23 (33.756)
  Social Limitations; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Social Limitations; Week 48;n=11, 27 | -20.20 (27.585) | -17.70 (27.087)
  Personal Relationships; Week 12;n=91, 79: number analyzed (Participants) | 91 | 79
  Personal Relationships; Week 12;n=91, 79 | -3.85 (21.528) | -5.06 (23.167)
  Personal Relationships; Week 24;n=13, 35: number analyzed (Participants) | 13 | 35
  Personal Relationships; Week 24;n=13, 35 | -10.26 (23.113) | -15.24 (30.883)
  Personal Relationships; Week 36;n=8, 20: number analyzed (Participants) | 8 | 20
  Personal Relationships; Week 36;n=8, 20 | -22.92 (30.780) | -15.00 (28.562)
  Personal Relationships; Week 48;n=8, 15: number analyzed (Participants) | 8 | 15
  Personal Relationships; Week 48;n=8, 15 | -22.92 (30.780) | -13.33 (23.738)
  Emotions; Week 12;n=122, 123: number analyzed (Participants) | 122 | 123
  Emotions; Week 12;n=122, 123 | -4.46 (22.841) | -14.63 (28.922)
  Emotions; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Emotions; Week 24;n=17, 54 | -22.22 (21.155) | -27.98 (30.198)
  Emotions; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Emotions; Week 36;n=12, 32 | -22.22 (21.711) | -23.26 (20.616)
  Emotions; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Emotions; Week 48;n=11, 27 | -20.20 (26.675) | -20.58 (28.362)
  Sleep/Energy; Week 12;n=122, 123: number analyzed (Participants) | 122 | 123
  Sleep/Energy; Week 12;n=122, 123 | 0.41 (23.223) | -12.74 (25.792)
  Sleep/Energy; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Sleep/Energy; Week 24;n=17, 54 | -13.73 (30.752) | -17.28 (26.886)
  Sleep/Energy; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Sleep/Energy; Week 36;n=12, 32 | -19.44 (23.391) | -11.98 (27.835)
  Sleep/Energy; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Sleep/Energy; Week 48;n=11, 27 | -16.67 (24.721) | -9.88 (28.592)
  Severity/Coping Measures; Week 12;n=122, 123: number analyzed (Participants) | 122 | 123
  Severity/Coping Measures; Week 12;n=122, 123 | -2.08 (16.950) | -11.54 (26.032)
  Severity/Coping Measures; Week 24;n=17, 54: number analyzed (Participants) | 17 | 54
  Severity/Coping Measures; Week 24;n=17, 54 | -9.80 (19.020) | -18.27 (28.260)
  Severity/Coping Measures; Week 36;n=12, 32: number analyzed (Participants) | 12 | 32
  Severity/Coping Measures; Week 36;n=12, 32 | -23.89 (18.740) | -14.17 (24.466)
  Severity/Coping Measures; Week 48;n=11, 27: number analyzed (Participants) | 11 | 27
  Severity/Coping Measures; Week 48;n=11, 27 | -18.18 (19.112) | -6.67 (26.667)

60. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Change From Baseline in KHQ Domain Scores
Description: KHQ is a 21 item questionnaire, consisting of 9 domains: GH (1[Very good] to 5[Very poor]), Int Imp (1[Not at all] to 4[A lot]), RL (1[Not at all] to 4[A lot]), PL (1[Not at all] to 4[A lot]), SL (0[not applicable] to 4[A lot]), PR (0[Not applicable] to 4[A lot]), Emotions (1[Not at all] to 4[Very much]), S/ E (1[Never] to 4[All the time]) and S/ C (1[Never] to 4[All the time]). Domain score for GH was calculated as score of one item minus 1/4x100; Int Imp: score of one item minus 1/3x100; RL, PL, PR, S/ E: summed scores of 2 items minus 2/6x100; SL, Emotions: summed scores of 3 items minus 3/9x100; S/ C: summed scores of 5 items minus 5/15x100. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 12, Week 24 and Week 36 in Treatment Cycle 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Scores on a scale
  General Health Perception; Week 0;n=108,88 | 8.1 (24.84) | 2.3 (23.86)
  General Health Perception; Week 12;n=106,85: number analyzed (Participants) | 106 | 85
  General Health Perception; Week 12;n=106,85 | -0.2 (25.47) | 2.6 (25.30)
  General Health Perception; Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  General Health Perception; Week 24;n=47,22 | 3.2 (27.39) | 2.3 (24.29)
  General Health Perception; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  General Health Perception; Week 36;n=25,8 | 1.0 (27.46) | 6.3 (29.12)
  Incontinence Impact; Week 0;n=108,88 | -2.78 (26.229) | -11.74 (31.171)
  Incontinence Impact; Week 12;n=106,85: number analyzed (Participants) | 106 | 85
  Incontinence Impact; Week 12;n=106,85 | -35.22 (35.584) | -23.14 (34.512)
  Incontinence Impact; Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  Incontinence Impact; Week 24;n=47,22 | -39.72 (35.193) | -36.36 (30.704)
  Incontinence Impact; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Incontinence Impact; Week 36;n=25,8 | -38.67 (38.103) | -37.50 (41.547)
  Role Limitations; Week 0;n= 107,88: number analyzed (Participants) | 107 | 88
  Role Limitations; Week 0;n= 107,88 | -0.31 (23.789) | -7.39 (25.753)
  Role Limitations; Week 12;n= 105,85: number analyzed (Participants) | 105 | 85
  Role Limitations; Week 12;n= 105,85 | -24.44 (33.178) | -22.35 (28.701)
  Role Limitations; Week 24;n=46,22: number analyzed (Participants) | 46 | 22
  Role Limitations; Week 24;n=46,22 | -27.17 (31.497) | -26.52 (33.198)
  Role Limitations; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Role Limitations; Week 36;n=25,8 | -30.67 (32.872) | -35.42 (38.253)
  Physical Limitations; Week 0;n=107,88: number analyzed (Participants) | 107 | 88
  Physical Limitations; Week 0;n=107,88 | 0.31 (25.181) | -4.73 (31.859)
  Physical Limitations; Week 12;n=105,85: number analyzed (Participants) | 105 | 85
  Physical Limitations; Week 12;n=105,85 | -24.76 (33.422) | -15.88 (30.851)
  Physical Limitations; Week 24;n=46,22: number analyzed (Participants) | 46 | 22
  Physical Limitations; Week 24;n=46,22 | -23.19 (37.594) | -17.42 (38.654)
  Physical Limitations; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Physical Limitations; Week 36;n=25,8 | -28.67 (34.534) | -31.25 (35.003)
  Social Limitations; Week 0;n=107,88: number analyzed (Participants) | 107 | 88
  Social Limitations; Week 0;n=107,88 | 2.96 (24.340) | -4.23 (27.733)
  Social Limitations; Week 12;n=105,85: number analyzed (Participants) | 105 | 85
  Social Limitations; Week 12;n=105,85 | -17.67 (31.283) | -9.35 (28.845)
  Social Limitations; Week 24;n=46,22: number analyzed (Participants) | 46 | 22
  Social Limitations; Week 24;n=46,22 | -17.51 (35.136) | -9.09 (35.368)
  Social Limitations; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Social Limitations; Week 36;n=25,8 | -22.00 (33.120) | -23.61 (21.771)
  Personal Relationships; Week 0;n=80,57: number analyzed (Participants) | 80 | 57
  Personal Relationships; Week 0;n=80,57 | -1.04 (20.600) | -2.63 (23.944)
  Personal Relationships; Week 12;n=79,54: number analyzed (Participants) | 79 | 54
  Personal Relationships; Week 12;n=79,54 | -6.75 (24.390) | -4.63 (26.385)
  Personal Relationships; Week 24;n=33,17: number analyzed (Participants) | 33 | 17
  Personal Relationships; Week 24;n=33,17 | -8.59 (27.677) | -14.71 (18.524)
  Personal Relationships; Week 36;n=19,6: number analyzed (Participants) | 19 | 6
  Personal Relationships; Week 36;n=19,6 | -7.02 (32.544) | -11.11 (13.608)
  Emotions; Week 0;n=108,88 | -2.67 (22.881) | -8.08 (26.192)
  Emotions; Week 12;n=106,85: number analyzed (Participants) | 106 | 85
  Emotions; Week 12;n=106,85 | -27.88 (29.347) | -14.64 (28.131)
  Emotions; Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  Emotions; Week 24;n=47,22 | -28.84 (31.653) | -18.69 (29.574)
  Emotions; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Emotions; Week 36;n=25,8 | -39.11 (29.766) | -18.06 (25.845)
  Sleep/Energy; Week 0;n=108,88 | 3.40 (22.986) | -8.90 (24.753)
  Sleep/Energy; Week 12;n=106,85: number analyzed (Participants) | 106 | 85
  Sleep/Energy; Week 12;n=106,85 | -14.31 (30.030) | -13.92 (25.569)
  Sleep/Energy; Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  Sleep/Energy; Week 24;n=47,22 | -11.70 (30.676) | -21.97 (22.647)
  Sleep/Energy; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Sleep/Energy; Week 36;n=25,8 | -13.33 (27.639) | -12.50 (24.801)
  Severity/Coping Measures; Week 0;n=108,88 | 0.56 (14.757) | -5.61 (23.573)
  Severity/Coping Measures; Week 12;n=106,85: number analyzed (Participants) | 106 | 85
  Severity/Coping Measures; Week 12;n=106,85 | -16.23 (25.845) | -11.37 (21.938)
  Severity/Coping Measures; Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  Severity/Coping Measures; Week 24;n=47,22 | -18.01 (28.041) | -16.97 (17.785)
  Severity/Coping Measures; Week 36;n=25,8: number analyzed (Participants) | 25 | 8
  Severity/Coping Measures; Week 36;n=25,8 | -19.20 (31.465) | -16.67 (28.284)

61. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Change From Baseline in KHQ Domain Scores
Description: as for outcome 60
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 12 and Week 24 in Treatment Cycle 3
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Treatment Cycle 3 Placebo / GSK1358820 100 U: Participants received a single (double-blind) treatment with Placebo (20 injections of 0.5 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received GSK1358820 100 U in Treatment Phase 2 (Treatment Cycle 3).
Arm/Group | Treatment Cycle 3 Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Scores on a scale
  General Health Perception; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  General Health Perception; Week 0;n=55,43 | 3.6 (22.27) | 6.4 (26.78)
  General Health Perception; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  General Health Perception; Week 12;n=54,42 | -3.2 (19.45) | -2.4 (29.64)
  General Health Perception; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  General Health Perception; Week 24;n=2,7 | 37.5 (17.68) | -7.1 (53.45)
  Incontinence Impact; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Incontinence Impact; Week 0;n=55,43 | -24.24 (32.365) | -10.08 (32.962)
  Incontinence Impact; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Incontinence Impact; Week 12;n=54,42 | -34.57 (29.647) | -16.67 (36.994)
  Incontinence Impact; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Incontinence Impact; Week 24;n=2,7 | 0.00 (0.000) | -14.29 (26.227)
  Role Limitations; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Role Limitations; Week 0;n=55,43 | -16.67 (26.058) | -15.12 (27.892)
  Role Limitations; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Role Limitations; Week 12;n=54,42 | -25.62 (33.912) | -10.32 (28.023)
  Role Limitations; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Role Limitations; Week 24;n=2,7 | 0.00 (0.000) | -7.14 (28.637)
  Physical Limitations; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Physical Limitations; Week 0;n=55,43 | -19.09 (27.670) | -13.95 (29.531)
  Physical Limitations; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Physical Limitations; Week 12;n=54,42 | -29.32 (29.662) | -12.70 (32.050)
  Physical Limitations; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Physical Limitations; Week 24;n=2,7 | 0.00 (0.000) | -28.57 (39.340)
  Social Limitations; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Social Limitations; Week 0;n=55,43 | -17.68 (24.195) | -6.07 (24.899)
  Social Limitations; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Social Limitations; Week 12;n=54,42 | -21.91 (28.724) | -7.54 (26.311)
  Social Limitations; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Social Limitations; Week 24;n=2,7 | -5.56 (7.857) | -7.94 (19.994)
  Personal Relationships; Week 0;n=42,23: number analyzed (Participants) | 42 | 23
  Personal Relationships; Week 0;n=42,23 | -7.14 (16.926) | 2.90 (17.875)
  Personal Relationships; Week 12;n=40,24: number analyzed (Participants) | 40 | 24
  Personal Relationships; Week 12;n=40,24 | -9.58 (19.203) | 4.17 (18.553)
  Personal Relationships; Week 24;n=1,4: number analyzed (Participants) | 1 | 4
  Personal Relationships; Week 24;n=1,4 | -16.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 16.67 (56.108)
  Emotions; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Emotions; Week 0;n=55,43 | -19.39 (22.551) | -10.08 (28.772)
  Emotions; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Emotions; Week 12;n=54,42 | -27.98 (28.776) | -8.47 (26.749)
  Emotions; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Emotions; Week 24;n=2,7 | -22.22 (15.713) | -7.94 (21.956)
  Sleep/Energy; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Sleep/Energy; Week 0;n=55,43 | -10.61 (22.536) | -7.75 (24.760)
  Sleep/Energy; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Sleep/Energy; Week 12;n=54,42 | -17.28 (26.095) | -10.71 (25.720)
  Sleep/Energy; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Sleep/Energy; Week 24;n=2,7 | -25.00 (11.785) | -7.14 (26.972)
  Severity/Coping Measures; Week 0;n=55,43: number analyzed (Participants) | 55 | 43
  Severity/Coping Measures; Week 0;n=55,43 | -11.15 (18.417) | -2.02 (17.429)
  Severity/Coping Measures; Week 12;n=54,42: number analyzed (Participants) | 54 | 42
  Severity/Coping Measures; Week 12;n=54,42 | -16.67 (20.992) | -4.76 (23.013)
  Severity/Coping Measures; Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Severity/Coping Measures; Week 24;n=2,7 | -6.67 (9.428) | -3.81 (18.402)

62. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Percentage of Participants With Positive Response on the Treatment Benefit Scale (TBS)
Description: Treatment benefit of GSK1358820 was assessed with TBS ranging from 1(Greatly improved) to 4 (Worsened). This questionnaire consists of 4 answers to 1 question by considering current condition of participants (urinary problems, urinary incontinence) compared to condition before participants received any study treatment in this trial. Positive treatment response was defined as score of either 1 or 2 (representing 'greatly improved' or 'improved').
Time Frame: Week 2, Week 6, Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Percentage of participants
  Week 2; n=124 ,124 | 22 | 60
  Week 6; n=124 ,124 | 23 | 64
  Week 12; n=124 ,124 | 17 | 57
  Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  Week 24; n=17, 54 | 53 | 69
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | 67 | 69
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | 45 | 70

63. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Percentage of Participants With Positive Response on the TBS
Description: as for outcome 62
Time Frame: Week 0, Week 2, Week 6, Week 12, Week 24 and Week 36 in Treatment Cycle 2
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Percentage of participants
  Week 0; n=108,88 | 7 | 40
  Week 2; n=108,86: number analyzed (Participants) | 108 | 86
  Week 2; n=108,86 | 81 | 70
  Week 6; n=108,86: number analyzed (Participants) | 108 | 86
  Week 6; n=108,86 | 79 | 69
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | 73 | 64
  Week 24; n=47,22: number analyzed (Participants) | 47 | 22
  Week 24; n=47,22 | 72 | 55
  Week 36; n=25,8: number analyzed (Participants) | 25 | 8
  Week 36; n=25,8 | 68 | 38

64. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Percentage of Participants With Positive Response on the TBS
Description: as for outcome 62
Time Frame: Week 0, Week 2, Week 6, Week 12 and Week 24 in Treatment Cycle 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Percentage of participants
  Week 0; n=56,43 | 61 | 49
  Week 2; n=56,43 | 64 | 60
  Week 6; n=55,43: number analyzed (Participants) | 55 | 43
  Week 6; n=55,43 | 65 | 63
  Week 12; n=54,42: number analyzed (Participants) | 54 | 42
  Week 12; n=54,42 | 63 | 55
  Week 24; n=2,7: number analyzed (Participants) | 2 | 7
  Week 24; n=2,7 | 0 | 29

65. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Changes From Baseline in Overactive Bladder Symptom Score (OABSS) Total Score
Description: Symptoms of frequency, nocturia, urinary urgency, and urge incontinence were assessed. OABSS questionnaire consisted of 4 questions: number of times participants urinate from waking in the morning until sleeping at night, ranging from 0 (<=7 times) to 1 (>=15 times); number of times participants wake up to urinate from sleeping at night until waking in the morning, ranging from 0 (0 times) to 3 (>=3 times); number of times for sudden desire to urinate, ranging from 0 (Not at all) to 5 (5 times a day or more); number of times of urine leakage, ranging from 0 (Not at all) to 5 (5 times a day or more). OABSS total score was calculated as the sum of scores for above 4 questions. The range of total score of OABSS was 0 to 15 with higher score indicating, more severity of symptoms. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Scores on a scale
  Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; n=122, 123 | -0.7 (2.05) | -3.4 (3.50)
  Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  Week 24; n=17, 54 | -2.7 (2.80) | -4.4 (3.32)
  Week 36; n=12 ,32: number analyzed (Participants) | 12 | 32
  Week 36; n=12 ,32 | -3.5 (2.02) | -3.9 (3.26)
  Week 48; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 48; n=11, 27 | -2.8 (2.68) | -3.3 (3.02)

66. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2): Changes From Baseline in OABSS Total Score
Description: as for outcome 65
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 12, Week 24 and Week 36 in Treatment Cycle 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 88
Scores on a scale
  Week 0; n=108,88 | -0.2 (1.78) | -1.5 (2.15)
  Week 12; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; n=106,85 | -4.1 (3.73) | -3.0 (2.89)
  Week 24;n=47,22: number analyzed (Participants) | 47 | 22
  Week 24;n=47,22 | -5.1 (3.62) | -3.3 (2.78)
  Week 36; n=25,8: number analyzed (Participants) | 25 | 8
  Week 36; n=25,8 | -5.1 (4.04) | -3.9 (3.48)

67. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3): Changes From Baseline in OABSS Total Score
Description: as for outcome 65
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 12 and Week 24 in Treatment Cycle 3
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 56 | 43
Scores on a scale
  Week 0; n=55,43: number analyzed (Participants) | 55 | 43
  Week 0; n=55,43 | -1.8 (1.93) | -1.5 (1.72)
  Week 12; n=54,42: number analyzed (Participants) | 54 | 42
  Week 12; n=54,42 | -3.2 (3.29) | -2.6 (2.89)
  Week 24;n=2,7: number analyzed (Participants) | 2 | 7
  Week 24;n=2,7 | -2.0 (2.83) | -1.6 (1.27)

68. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or other situations as per medical or scientific judgment.
Time Frame: Up to 48 weeks in Treatment Cycle 1
Population: Safety for double blind phase (SPDB) Population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Any SAE | 6 | 8
  Any non-SAE | 29 | 53

69. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With SAEs and Non-SAEs: Placebo/GSK1358820 100 U
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or other situations as per medical or scientific judgment. Safety Population 1 comprised of all participants who received at least one dose of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Participants
  Any SAE | 5
  Any non-SAE | 49

70. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With SAEs and Non-SAEs: GSK1358820 100 U/GSK1358820 100 U
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or other situations as per medical or scientific judgment. Safety Population 2 comprised of all participants who received at least two doses of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 88
Participants
  Any SAE | 5
  Any non-SAE | 40

71. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With SAEs and Non-SAEs: Placebo/GSK1358820 100 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 56
Participants
  Any SAE | 0
  Any non-SAE | 22

72. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With SAEs and Non-SAEs: GSK1358820 100 U/GSK1358820 100 U
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or other situations as per medical or scientific judgment. Safety Population 3 comprised of all participants who received at least three doses of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 43
Participants
  Any SAE | 1
  Any non-SAE | 19

73. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in seated position after 5 minutes rest for participants at indicated time points. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at specified time point were analyzed (represented by n=X) in category titles.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Millimeter of mercury
  SBP; Week 2; n=124, 124 | -0.6 (13.24) | -1.5 (13.17)
  SBP; Week 6; n=124, 123: number analyzed (Participants) | 124 | 123
  SBP; Week 6; n=124, 123 | -2.8 (13.00) | -1.1 (14.47)
  SBP; Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  SBP; Week 12; n=122, 123 | -2.9 (14.05) | -1.6 (14.42)
  SBP; Week 18; n=23, 65: number analyzed (Participants) | 23 | 65
  SBP; Week 18; n=23, 65 | 0.3 (19.61) | -5.8 (14.17)
  SBP; Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  SBP; Week 24; n=17, 54 | -4.8 (18.70) | -5.2 (14.53)
  SBP; Week 30; n=14, 47: number analyzed (Participants) | 14 | 47
  SBP; Week 30; n=14, 47 | -2.6 (23.22) | -4.6 (14.85)
  SBP; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  SBP; Week 36; n=12, 32 | -8.5 (18.02) | -5.2 (15.94)
  SBP; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  SBP; Week 42; n=11, 27 | -6.1 (20.53) | -5.8 (16.69)
  SBP; Week 48; n=16, 36: number analyzed (Participants) | 16 | 36
  SBP; Week 48; n=16, 36 | 4.5 (13.85) | -1.5 (16.48)
  DBP; Week 2; n=124, 124 | 0.2 (9.39) | -1.4 (9.43)
  DBP; Week 6; n=124, 123: number analyzed (Participants) | 124 | 123
  DBP; Week 6; n=124, 123 | -1.6 (10.03) | 0.1 (10.79)
  DBP; Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  DBP; Week 12; n=122, 123 | -1.8 (10.89) | -1.6 (10.48)
  DBP; Week 18; n=23, 65: number analyzed (Participants) | 23 | 65
  DBP; Week 18; n=23, 65 | -1.5 (11.61) | -3.0 (8.89)
  DBP; Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  DBP; Week 24; n=17, 54 | -5.0 (8.85) | -3.1 (11.46)
  DBP; Week 30; n=14, 47: number analyzed (Participants) | 14 | 47
  DBP; Week 30; n=14, 47 | -1.4 (9.44) | -2.1 (10.97)
  DBP; Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  DBP; Week 36; n=12, 32 | -4.9 (7.88) | -4.3 (12.08)
  DBP; Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  DBP; Week 42; n=11, 27 | -4.7 (10.03) | -4.1 (12.05)
  DBP; Week 48; n=16, 36: number analyzed (Participants) | 16 | 36
  DBP; Week 48; n=16, 36 | 0.3 (6.56) | -2.2 (12.79)

74. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in SBP and DBP: Placebo/GSK1358820 100 U
Description: as for outcome 73
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at specified time point were analyzed (represented by n=X) in category titles.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Millimeter of mercury
  SBP; Week 0; n=107: number analyzed (Participants) | 107
  SBP; Week 0; n=107 | -1.4 (14.54)
  SBP; Week 2; n=108 | -2.0 (14.11)
  SBP; Week 6; n=108 | -2.9 (13.70)
  SBP; Week 12; n=106: number analyzed (Participants) | 106
  SBP; Week 12; n=106 | -0.8 (13.40)
  SBP; Week 18; n=82: number analyzed (Participants) | 82
  SBP; Week 18; n=82 | -2.6 (14.06)
  SBP; Week 24; n=45: number analyzed (Participants) | 45
  SBP; Week 24; n=45 | -1.4 (14.51)
  SBP; Week 30; n=37: number analyzed (Participants) | 37
  SBP; Week 30; n=37 | -2.8 (15.56)
  SBP; Week 36; n=7: number analyzed (Participants) | 7
  SBP; Week 36; n=7 | -1.9 (13.46)
  SBP; Week 48; n=52: number analyzed (Participants) | 52
  SBP; Week 48; n=52 | -1.4 (14.03)
  DBP; Week 0; n=107: number analyzed (Participants) | 107
  DBP; Week 0; n=107 | -0.7 (10.38)
  DBP; Week 2; n=108 | -0.7 (10.65)
  DBP; Week 6; n=108 | -1.5 (11.43)
  DBP; Week 12; n=106: number analyzed (Participants) | 106
  DBP; Week 12; n=106 | -1.5 (11.19)
  DBP; Week 18; n=82: number analyzed (Participants) | 82
  DBP; Week 18; n=82 | -1.6 (11.30)
  DBP; Week 24; n=45: number analyzed (Participants) | 45
  DBP; Week 24; n=45 | -1.8 (9.73)
  DBP; Week 30; n=37: number analyzed (Participants) | 37
  DBP; Week 30; n=37 | -1.3 (9.23)
  DBP; Week 36; n=7: number analyzed (Participants) | 7
  DBP; Week 36; n=7 | 1.6 (7.18)
  DBP; Week 48; n=52: number analyzed (Participants) | 52
  DBP; Week 48; n=52 | -0.2 (8.30)

75. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in SBP and DBP: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 73
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. All the participants in this population were analyzed (124 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Millimeter of mercury
  SBP; Week 0; n=87: number analyzed (Participants) | 87
  SBP; Week 0; n=87 | -1.6 (12.72)
  SBP; Week 2; n=87: number analyzed (Participants) | 87
  SBP; Week 2; n=87 | -1.1 (15.93)
  SBP; Week 6; n=86: number analyzed (Participants) | 86
  SBP; Week 6; n=86 | -3.8 (16.05)
  SBP; Week 12; n=85: number analyzed (Participants) | 85
  SBP; Week 12; n=85 | -2.8 (13.94)
  SBP; Week 18; n=39: number analyzed (Participants) | 39
  SBP; Week 18; n=39 | -8.3 (12.85)
  SBP; Week 24; n=19: number analyzed (Participants) | 19
  SBP; Week 24; n=19 | 1.2 (18.38)
  SBP; Week 30; n=14: number analyzed (Participants) | 14
  SBP; Week 30; n=14 | 0.6 (10.80)
  SBP; Week 48; n=45: number analyzed (Participants) | 45
  SBP; Week 48; n=45 | -1.8 (16.33)
  DBP; Week 0; n=87: number analyzed (Participants) | 87
  DBP; Week 0; n=87 | -1.3 (9.59)
  DBP; Week 2; n=87: number analyzed (Participants) | 87
  DBP; Week 2; n=87 | -0.6 (10.17)
  DBP; Week 6; n=86: number analyzed (Participants) | 86
  DBP; Week 6; n=86 | -2.6 (11.67)
  DBP; Week 12; n=85: number analyzed (Participants) | 85
  DBP; Week 12; n=85 | -2.5 (10.55)
  DBP; Week 18; n=39: number analyzed (Participants) | 39
  DBP; Week 18; n=39 | -6.3 (9.93)
  DBP; Week 24; n=19: number analyzed (Participants) | 19
  DBP; Week 24; n=19 | -2.3 (11.57)
  DBP; Week 30; n=14: number analyzed (Participants) | 14
  DBP; Week 30; n=14 | -0.9 (9.53)
  DBP; Week 48; n=45: number analyzed (Participants) | 45
  DBP; Week 48; n=45 | -2.2 (9.74)

76. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in SBP and DBP: Placebo/GSK1358820 100 U
Description: as for outcome 73
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 1. All the participants in this population were analyzed (108 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Millimeter of mercury
  SBP; Week 0; n=56: number analyzed (Participants) | 56
  SBP; Week 0; n=56 | -1.2 (14.48)
  SBP; Week 2; n=56: number analyzed (Participants) | 56
  SBP; Week 2; n=56 | -2.4 (12.28)
  SBP; Week 6; n=55: number analyzed (Participants) | 55
  SBP; Week 6; n=55 | -2.6 (15.91)
  SBP; Week 12; n=53: number analyzed (Participants) | 53
  SBP; Week 12; n=53 | -3.9 (17.70)
  SBP; Week 18; n=19: number analyzed (Participants) | 19
  SBP; Week 18; n=19 | -3.2 (12.08)
  SBP; Week 24; n=1: number analyzed (Participants) | 1
  SBP; Week 24; n=1 | -23.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SBP; Week 48; n=56: number analyzed (Participants) | 56
  SBP; Week 48; n=56 | -1.7 (13.58)
  DBP; Week 0; n=56: number analyzed (Participants) | 56
  DBP; Week 0; n=56 | -0.9 (10.19)
  DBP; Week 2; n=56: number analyzed (Participants) | 56
  DBP; Week 2; n=56 | -2.5 (11.61)
  DBP; Week 6; n=55: number analyzed (Participants) | 55
  DBP; Week 6; n=55 | -1.4 (13.08)
  DBP; Week 12; n=53: number analyzed (Participants) | 53
  DBP; Week 12; n=53 | -3.2 (11.76)
  DBP; Week 18; n=19: number analyzed (Participants) | 19
  DBP; Week 18; n=19 | -2.3 (13.23)
  DBP; Week 24; n=1: number analyzed (Participants) | 1
  DBP; Week 24; n=1 | -19.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  DBP; Week 48; n=56: number analyzed (Participants) | 56
  DBP; Week 48; n=56 | -2.8 (11.24)

77. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in SBP and DBP: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 73
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Millimeter of mercury
  SBP; Week 0; n=43: number analyzed (Participants) | 43
  SBP; Week 0; n=43 | -3.0 (15.49)
  SBP; Week 2; n=43: number analyzed (Participants) | 43
  SBP; Week 2; n=43 | -2.5 (16.00)
  SBP; Week 6; n=43: number analyzed (Participants) | 43
  SBP; Week 6; n=43 | -4.5 (15.85)
  SBP; Week 12; n=40: number analyzed (Participants) | 40
  SBP; Week 12; n=40 | -3.2 (17.50)
  SBP; Week 18; n=27: number analyzed (Participants) | 27
  SBP; Week 18; n=27 | -3.4 (13.58)
  SBP; Week 48; n=43: number analyzed (Participants) | 43
  SBP; Week 48; n=43 | -4.7 (14.62)
  DBP; Week 0; n=43: number analyzed (Participants) | 43
  DBP; Week 0; n=43 | -1.1 (10.21)
  DBP; Week 2; n=43: number analyzed (Participants) | 43
  DBP; Week 2; n=43 | -3.1 (10.68)
  DBP; Week 6; n=43: number analyzed (Participants) | 43
  DBP; Week 6; n=43 | -3.7 (10.08)
  DBP; Week 12; n=40: number analyzed (Participants) | 40
  DBP; Week 12; n=40 | -1.2 (10.21)
  DBP; Week 18; n=27: number analyzed (Participants) | 27
  DBP; Week 18; n=27 | -1.5 (7.65)
  DBP; Week 48; n=43: number analyzed (Participants) | 43
  DBP; Week 48; n=43 | -4.0 (10.95)

78. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Heart Rate
Description: Heart rate was measured in seated position after 5 minutes rest for participants at indicated time points. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1) and Week 2, Week 6, Week 12, Week 18, Week 24 Week 30, Week 36, Week 42 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Beats per minute
  Week 2; n=124, 124 | -2.2 (8.39) | -1.2 (10.62)
  Week 6; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 6; n=124, 123 | -2.7 (10.06) | -0.8 (10.56)
  Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; n=122, 123 | -3.8 (9.18) | -1.6 (10.36)
  Week 18; n=23, 65: number analyzed (Participants) | 23 | 65
  Week 18; n=23, 65 | -4.5 (10.39) | -3.8 (10.11)
  Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  Week 24; n=17, 54 | -6.6 (13.24) | -2.6 (10.98)
  Week 30; n=14, 47: number analyzed (Participants) | 14 | 47
  Week 30; n=14, 47 | -5.2 (7.68) | -2.7 (9.94)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -5.7 (8.58) | -3.4 (9.64)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | 2.3 (10.69) | -2.1 (9.79)
  Week 48; n=16, 36: number analyzed (Participants) | 16 | 36
  Week 48; n=16, 36 | -3.8 (8.69) | -3.6 (10.06)

79. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Heart Rate: Placebo/GSK1358820 100 U
Description: as for outcome 78
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24 Week 30, Week 36 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Beats per minute
  Week 0; n=107: number analyzed (Participants) | 107
  Week 0; n=107 | -0.4 (9.42)
  Week 2; n=108 | -1.8 (10.06)
  Week 6; n=108 | -1.4 (10.32)
  Week 12; n=106: number analyzed (Participants) | 106
  Week 12; n=106 | -4.3 (10.03)
  Week 18; n=82: number analyzed (Participants) | 82
  Week 18; n=82 | -4.1 (9.12)
  Week 24; n=45: number analyzed (Participants) | 45
  Week 24; n=45 | -0.9 (9.43)
  Week 30; n=37: number analyzed (Participants) | 37
  Week 30; n=37 | -0.7 (9.23)
  Week 36; n=7: number analyzed (Participants) | 7
  Week 36; n=7 | -0.6 (5.88)
  Week 48; n=52: number analyzed (Participants) | 52
  Week 48; n=52 | -3.2 (10.49)

80. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Heart Rate: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 78
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24 Week 30 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Beats per minute
  Week 0; n=87: number analyzed (Participants) | 87
  Week 0; n=87 | 1.9 (9.75)
  Week 2; n=87: number analyzed (Participants) | 87
  Week 2; n=87 | 0.6 (10.68)
  Week 6; n=86: number analyzed (Participants) | 86
  Week 6; n=86 | 1.6 (10.51)
  Week 12; n=85: number analyzed (Participants) | 85
  Week 12; n=85 | -1.8 (11.01)
  Week 18; n=39: number analyzed (Participants) | 39
  Week 18; n=39 | -0.0 (10.35)
  Week 24; n=19: number analyzed (Participants) | 19
  Week 24; n=19 | 0.3 (9.67)
  Week 30; n=14: number analyzed (Participants) | 14
  Week 30; n=14 | 2.7 (9.24)
  Week 48; n=45: number analyzed (Participants) | 45
  Week 48; n=45 | 1.0 (9.17)

81. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Heart Rate: Placebo/GSK1358820 100 U
Description: as for outcome 78
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Beats per minute
  Week 0; n=56: number analyzed (Participants) | 56
  Week 0; n=56 | 0.2 (9.28)
  Week 2; n=56: number analyzed (Participants) | 56
  Week 2; n=56 | -2.3 (9.26)
  Week 6; n=55: number analyzed (Participants) | 55
  Week 6; n=55 | -2.9 (9.24)
  Week 12; n=53: number analyzed (Participants) | 53
  Week 12; n=53 | -3.8 (10.28)
  Week 18; n=19: number analyzed (Participants) | 19
  Week 18; n=19 | -0.6 (11.08)
  Week 24; n=1: number analyzed (Participants) | 1
  Week 24; n=1 | 6.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 48; n=56: number analyzed (Participants) | 56
  Week 48; n=56 | -1.8 (11.47)

82. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Heart Rate: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 78
Time Frame: as for outcome 77
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Beats per minute
  Week 0; n=43: number analyzed (Participants) | 43
  Week 0; n=43 | 1.2 (12.33)
  Week 2; n=43: number analyzed (Participants) | 43
  Week 2; n=43 | -3.3 (9.69)
  Week 6; n=43: number analyzed (Participants) | 43
  Week 6; n=43 | -3.1 (10.19)
  Week 12; n=40: number analyzed (Participants) | 40
  Week 12; n=40 | -5.7 (10.99)
  Week 18; n=27: number analyzed (Participants) | 27
  Week 18; n=27 | -3.7 (11.57)
  Week 48; n=43: number analyzed (Participants) | 43
  Week 48; n=43 | -2.5 (11.20)

83. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in Temperature
Description: Temperature was measured in seated position after 5 minutes rest for participants at indicated time points. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 73
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Degree Celsius
  Week 2; n=124, 124 | -0.04 (0.403) | -0.02 (0.460)
  Week 6; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 6; n=124, 123 | -0.03 (0.452) | -0.03 (0.497)
  Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; n=122, 123 | -0.13 (0.501) | -0.04 (0.470)
  Week 18; n=23, 65: number analyzed (Participants) | 23 | 65
  Week 18; n=23, 65 | -0.28 (0.540) | -0.01 (0.571)
  Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  Week 24; n=17, 54 | -0.26 (0.433) | 0.06 (0.497)
  Week 30; n=14, 47: number analyzed (Participants) | 14 | 47
  Week 30; n=14, 47 | -0.17 (0.446) | 0.01 (0.450)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | -0.11 (0.318) | -0.03 (0.450)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -0.10 (0.436) | -0.03 (0.525)
  Week 48; n=16, 36: number analyzed (Participants) | 16 | 36
  Week 48; n=16, 36 | 0.05 (0.447) | -0.01 (0.467)

84. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Temperature: Placebo/GSK1358820 100 U
Description: as for outcome 83
Time Frame: as for outcome 74
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Degree Celsius
  Week 0; n=107: number analyzed (Participants) | 107
  Week 0; n=107 | 0.01 (0.505)
  Week 2; n=108 | -0.06 (0.485)
  Week 6; n=108 | -0.04 (0.433)
  Week 12; n=106: number analyzed (Participants) | 106
  Week 12; n=106 | -0.09 (0.446)
  Week 18; n=82: number analyzed (Participants) | 82
  Week 18; n=82 | -0.09 (0.469)
  Week 24; n=45: number analyzed (Participants) | 45
  Week 24; n=45 | -0.08 (0.526)
  Week 30; n=37: number analyzed (Participants) | 37
  Week 30; n=37 | -0.08 (0.458)
  Week 36; n=7: number analyzed (Participants) | 7
  Week 36; n=7 | 0.06 (0.526)
  Week 48; n=52: number analyzed (Participants) | 52
  Week 48; n=52 | -0.12 (0.478)

85. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Temperature: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 83
Time Frame: as for outcome 75
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Degree Celsius
  Week 0; n=87: number analyzed (Participants) | 87
  Week 0; n=87 | -0.01 (0.465)
  Week 2; n=87: number analyzed (Participants) | 87
  Week 2; n=87 | -0.02 (0.549)
  Week 6; n=86: number analyzed (Participants) | 86
  Week 6; n=86 | -0.02 (0.456)
  Week 12; n=85: number analyzed (Participants) | 85
  Week 12; n=85 | -0.02 (0.472)
  Week 18; n=39: number analyzed (Participants) | 39
  Week 18; n=39 | -0.02 (0.480)
  Week 24; n=19: number analyzed (Participants) | 19
  Week 24; n=19 | 0.02 (0.459)
  Week 30; n=14: number analyzed (Participants) | 14
  Week 30; n=14 | -0.01 (0.403)
  Week 48; n=45: number analyzed (Participants) | 45
  Week 48; n=45 | 0.02 (0.539)

86. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Temperature: Placebo/GSK1358820 100 U
Description: as for outcome 83
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Degree Celsius
  Week 0; n=56: number analyzed (Participants) | 56
  Week 0; n=56 | 0.07 (0.507)
  Week 2; n=56: number analyzed (Participants) | 56
  Week 2; n=56 | 0.01 (0.511)
  Week 6; n=55: number analyzed (Participants) | 55
  Week 6; n=55 | 0.02 (0.471)
  Week 12; n=53: number analyzed (Participants) | 53
  Week 12; n=53 | 0.01 (0.472)
  Week 18; n=19: number analyzed (Participants) | 19
  Week 18; n=19 | 0.02 (0.527)
  Week 24; n=1: number analyzed (Participants) | 1
  Week 24; n=1 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 48; n=56: number analyzed (Participants) | 56
  Week 48; n=56 | -0.04 (0.500)

87. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Temperature: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 83
Time Frame: as for outcome 77
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Degree Celsius
  Week 0; n=43: number analyzed (Participants) | 43
  Week 0; n=43 | -0.11 (0.429)
  Week 2; n=43: number analyzed (Participants) | 43
  Week 2; n=43 | -0.15 (0.502)
  Week 6; n=43: number analyzed (Participants) | 43
  Week 6; n=43 | -0.04 (0.530)
  Week 12; n=40: number analyzed (Participants) | 40
  Week 12; n=40 | -0.09 (0.471)
  Week 18; n=27: number analyzed (Participants) | 27
  Week 18; n=27 | -0.18 (0.481)
  Week 48; n=43: number analyzed (Participants) | 43
  Week 48; n=43 | -0.17 (0.447)

88. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Shift From Baseline Relative to Normal Range in Chemistry Results
Description: Blood samples were collected for analysis of following clinical chemistry parameters; Albumin, Alkaline Phosphatase (Alk Phosp), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Direct Bilirubin (Bil), Total Bil, Calcium, Chloride, Creatinine, Glucose, Potassium, Sodium, Total Protein (T Protein), Urea/blood urea nitrogen (BUN) and Uric acid. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, are recorded in the To Normal or No Change category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose on Day 1), Week 12 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: SPDB Population. All the participants in this population were analyzed (124, 124 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Week 12:Albumin; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Albumin; To Low; n=122, 122 | 0 | 1
  Week12:Albumin; To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Albumin; To Normal or No Change; n=122, 122 | 122 | 121
  Week12:Albumin; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Albumin; To High; n=122, 122 | 0 | 0
  Week 48:Albumin; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Albumin; To Low; n=16,36 | 0 | 1
  Week48:Albumin; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Albumin; To Normal or No Change; n=16,36 | 16 | 35
  Week48:Albumin; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Albumin; To High; n=16,36 | 0 | 0
  Week12:Alk Phosp; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Alk Phosp; To Low; n=122, 122 | 1 | 2
  Week12:Alk Phosp;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Alk Phosp;To Normal or No Change;n=122,122 | 116 | 117
  Week12:Alk Phosp; To High; n= 122 ,122: number analyzed (Participants) | 122 | 122
  Week12:Alk Phosp; To High; n= 122 ,122 | 5 | 3
  Week48:Alk Phosp; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Alk Phosp; To Low; n=16,36 | 0 | 1
  Week48:Alk Phosp;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Alk Phosp;To Normal or No Change;n=16,36 | 15 | 35
  Week48:Alk Phosp; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Alk Phosp; To High; n=16,36 | 1 | 0
  Week12:ALT;To Low; n= 122 ,122: number analyzed (Participants) | 122 | 122
  Week12:ALT;To Low; n= 122 ,122 | 0 | 0
  Week12:ALT;To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:ALT;To Normal or No Change; n=122, 122 | 120 | 117
  Week12:ALT; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:ALT; To High; n=122, 122 | 2 | 5
  Week48:ALT;To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:ALT;To Low; n=16,36 | 0 | 0
  Week48:ALT;To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:ALT;To Normal or No Change; n=16,36 | 16 | 36
  Week48:ALT; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:ALT; To High; n=16,36 | 0 | 0
  Week12:AST;To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:AST;To Low; n=122, 122 | 0 | 0
  Week12:AST; To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:AST; To Normal or No Change; n=122, 122 | 122 | 119
  Week12:AST; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:AST; To High; n=122, 122 | 0 | 3
  Week48:AST;To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:AST;To Low; n=16,36 | 0 | 0
  Week48:AST; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:AST; To Normal or No Change; n=16,36 | 16 | 35
  Week48:AST; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:AST; To High; n=16,36 | 0 | 1
  Week12:Direct Bil; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Direct Bil; To Low; n=122, 122 | 0 | 0
  Week12:Direct Bil;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Direct Bil;To Normal or No Change;n=122,122 | 122 | 122
  Week12:Direct Bil; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Direct Bil; To High; n=122, 122 | 0 | 0
  Week48:Direct Bil; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Direct Bil; To Low; n=16,36 | 0 | 0
  Week48:Direct Bil; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Direct Bil; To Normal or No Change; n=16,36 | 16 | 36
  Week48:Direct Bil; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Direct Bil; To High; n=16,36 | 0 | 0
  Week12:Total Bil; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Total Bil; To Low; n=122, 122 | 0 | 0
  Week12:Total Bil;To Normal or NoChange; n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Total Bil;To Normal or NoChange; n=122,122 | 120 | 121
  Week12:Total Bil; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Total Bil; To High; n=122, 122 | 2 | 1
  Week48:Total Bil; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Total Bil; To Low; n=16,36 | 0 | 0
  Week48:Total Bil; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Total Bil; To Normal or No Change; n=16,36 | 16 | 36
  Week48:Total Bil; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Total Bil; To High; n=16,36 | 0 | 0
  Week12:Calcium; To Low; n=122, 121: number analyzed (Participants) | 122 | 121
  Week12:Calcium; To Low; n=122, 121 | 5 | 4
  Week12:Calcium; To Normal or No Change; n=122, 121: number analyzed (Participants) | 122 | 121
  Week12:Calcium; To Normal or No Change; n=122, 121 | 117 | 117
  Week12:Calcium; To High; n=122, 121: number analyzed (Participants) | 122 | 121
  Week12:Calcium; To High; n=122, 121 | 0 | 0
  Week48:Calcium; To Low; n=16,35: number analyzed (Participants) | 16 | 35
  Week48:Calcium; To Low; n=16,35 | 1 | 3
  Week48:Calcium; To Normal or No Change; n=16,35: number analyzed (Participants) | 16 | 35
  Week48:Calcium; To Normal or No Change; n=16,35 | 15 | 32
  Week48:Calcium; To High; n=16,35: number analyzed (Participants) | 16 | 35
  Week48:Calcium; To High; n=16,35 | 0 | 0
  Week12:Chloride; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Chloride; To Low; n=122, 122 | 0 | 2
  Week12:Chloride; To Normal or No Change; n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Chloride; To Normal or No Change; n=122,122 | 121 | 119
  Week12:Chloride; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Chloride; To High; n=122, 122 | 1 | 1
  Week48:Chloride; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Chloride; To Low; n=16,36 | 0 | 1
  Week48:Chloride; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Chloride; To Normal or No Change; n=16,36 | 16 | 34
  Week48:Chloride; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Chloride; To High; n=16,36 | 0 | 1
  Week12:Creatinine; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Creatinine; To Low; n=122, 122 | 4 | 3
  Week12:Creatinine;To Normal or NoChange; n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Creatinine;To Normal or NoChange; n=122,122 | 114 | 116
  Week12:Creatinine; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Creatinine; To High; n=122, 122 | 4 | 3
  Week48:Creatinine; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Creatinine; To Low; n=16,36 | 0 | 0
  Week48:Creatinine; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Creatinine; To Normal or No Change; n=16,36 | 16 | 36
  Week48:Creatinine; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Creatinine; To High; n=16,36 | 0 | 0
  Week12:Glucose; To Low; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:Glucose; To Low; n=122, 123 | 1 | 0
  Week12:Glucose; To Normal or No Change; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:Glucose; To Normal or No Change; n=122, 123 | 101 | 106
  Week12:Glucose; To High; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:Glucose; To High; n=122, 123 | 20 | 17
  Week48:Glucose; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Glucose; To Low; n=16,36 | 0 | 0
  Week48:Glucose; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Glucose; To Normal or No Change; n=16,36 | 15 | 31
  Week48:Glucose; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Glucose; To High; n=16,36 | 1 | 5
  Week12:Potassium; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Potassium; To Low; n=122, 122 | 1 | 3
  Week12:Potassium;To Normal or No Change; n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Potassium;To Normal or No Change; n=122,122 | 121 | 118
  Week12:Potassium; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Potassium; To High; n=122, 122 | 0 | 1
  Week48:Potassium; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Potassium; To Low; n=16,36 | 1 | 0
  Week48:Potassium; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Potassium; To Normal or No Change; n=16,36 | 15 | 36
  Week48:Potassium; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Potassium; To High; n=16,36 | 0 | 0
  Week12:Sodium; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Sodium; To Low; n=122, 122 | 0 | 5
  Week12:Sodium;To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Sodium;To Normal or No Change; n=122, 122 | 122 | 116
  Week12:Sodium; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Sodium; To High; n=122, 122 | 0 | 1
  Week48:Sodium; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Sodium; To Low; n=16,36 | 0 | 3
  Week48:Sodium;To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Sodium;To Normal or No Change; n=16,36 | 16 | 32
  Week48:Sodium; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Sodium; To High; n=16,36 | 0 | 1
  Week12:T Protein; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:T Protein; To Low; n=122, 122 | 14 | 14
  Week12: T Protein;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12: T Protein;To Normal or No Change;n=122,122 | 108 | 108
  Week12:T Protein; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:T Protein; To High; n=122, 122 | 0 | 0
  Week48:T Protein; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Protein; To Low; n=16,36 | 1 | 5
  Week48:T Protein;To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Protein;To Normal or No Change; n=16,36 | 15 | 31
  Week48:T Protein; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Protein; To High; n=16,36 | 0 | 0
  Week12:Urea/BUN; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Urea/BUN; To Low; n=122, 122 | 1 | 1
  Week12Urea/BUN; To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12Urea/BUN; To Normal or No Change; n=122, 122 | 119 | 116
  Week12:Urea/BUN; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Urea/BUN; To High; n=122, 122 | 2 | 5
  Week48:Urea/BUN; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Urea/BUN; To Low; n=16,36 | 0 | 0
  Week48:Urea/BUN; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Urea/BUN; To Normal or No Change; n=16,36 | 16 | 35
  Week48:Urea/BUN; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Urea/BUN; To High; n=16,36 | 0 | 1
  Week12:Uric acid; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Uric acid; To Low; n=122, 122 | 1 | 2
  Week12:Uric acid;To Normal or No Change;n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Uric acid;To Normal or No Change;n=122, 122 | 116 | 117
  Week12:Uric acid; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Uric acid; To High; n=122, 122 | 5 | 3
  Week48:Uric acid; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Uric acid; To Low; n=16,36 | 0 | 1
  Week48:Uric acid;To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Uric acid;To Normal or No Change; n=16,36 | 16 | 34
  Week48:Uric acid; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Uric acid; To High; n=16,36 | 0 | 1

89. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Shift From Baseline Relative to Normal Range in Chemistry Results
Description: Blood samples were collected for analysis of following clinical chemistry parameters; Albumin, Alk Phosp, ALT, AST, Direct Bil, Total Bil, Calcium, Chloride, Creatinine, Glucose, Potassium, Sodium, T Protein, Urea/BUN and Uric acid. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, are recorded in the To Normal or No Change category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. All the participants in this population were analyzed (108, 124 participants) but only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week 12:Albumin; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Albumin; To Low; n=106,85 | 3 | 0
  Week12:Albumin; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Albumin; To Normal or No Change; n=106,85 | 103 | 85
  Week12:Albumin; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Albumin; To High; n=106,85 | 0 | 0
  Week 48:Albumin; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48:Albumin; To Low; n=52,45 | 0 | 1
  Week48:Albumin; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Albumin; To Normal or No Change; n=52,45 | 52 | 44
  Week48:Albumin; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Albumin; To High; n=52,45 | 0 | 0
  Week12:Alk Phosp; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Alk Phosp; To Low; n=106,85 | 1 | 0
  Week12:Alk Phosp;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Alk Phosp;To Normal or No Change;n=106,85 | 98 | 81
  Week12:Alk Phosp; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Alk Phosp; To High; n=106,85 | 7 | 4
  Week48:Alk Phosp; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Alk Phosp; To Low; n=52,45 | 0 | 0
  Week48:Alk Phosp;To Normal or No Change;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Alk Phosp;To Normal or No Change;n=52,45 | 49 | 43
  Week48:Alk Phosp; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Alk Phosp; To High; n=52,45 | 3 | 2
  Week12:ALT;To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:ALT;To Low; n=106,85 | 0 | 0
  Week12:ALT;To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:ALT;To Normal or No Change; n=106,85 | 104 | 83
  Week12:ALT; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:ALT; To High; n=106,85 | 2 | 2
  Week48:ALT;To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:ALT;To Low; n=52,45 | 0 | 0
  Week48:ALT;To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:ALT;To Normal or No Change; n=52,45 | 50 | 42
  Week48:ALT; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:ALT; To High; n=52,45 | 2 | 3
  Week12:AST;To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:AST;To Low; n=106,85 | 0 | 0
  Week12:AST; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:AST; To Normal or No Change; n=106,85 | 103 | 83
  Week12:AST; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:AST; To High; n=106,85 | 3 | 2
  Week48:AST;To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:AST;To Low; n=52,45 | 0 | 0
  Week48:AST; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:AST; To Normal or No Change; n=52,45 | 50 | 42
  Week48:AST; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:AST; To High; n=52,45 | 2 | 3
  Week12:Direct Bil; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Direct Bil; To Low; n=106,85 | 0 | 0
  Week12:Direct Bil;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Direct Bil;To Normal or No Change;n=106,85 | 106 | 84
  Week12:Direct Bil; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Direct Bil; To High; n=106,85 | 0 | 1
  Week48:Direct Bil; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Direct Bil; To Low; n=52,45 | 0 | 0
  Week48:Direct Bil; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Direct Bil; To Normal or No Change; n=52,45 | 52 | 45
  Week48:Direct Bil; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Direct Bil; To High; n=52,45 | 0 | 0
  Week12:Total Bil; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Total Bil; To Low; n=106,85 | 0 | 0
  Week12:Total Bil;To Normal or NoChange; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Total Bil;To Normal or NoChange; n=106,85 | 104 | 84
  Week12:Total Bil; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Total Bil; To High; n=106,85 | 2 | 1
  Week48:Total Bil; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Total Bil; To Low; n=52,45 | 0 | 0
  Week48:Total Bil; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Total Bil; To Normal or No Change; n=52,45 | 52 | 43
  Week48:Total Bil; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Total Bil; To High; n=52,45 | 0 | 2
  Week12:Calcium; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Calcium; To Low; n=106,85 | 1 | 1
  Week12:Calcium; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Calcium; To Normal or No Change; n=106,85 | 105 | 84
  Week12:Calcium; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Calcium; To High; n=106,85 | 0 | 0
  Week48:Calcium; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Calcium; To Low; n=52,45 | 1 | 1
  Week48:Calcium; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Calcium; To Normal or No Change; n=52,45 | 51 | 44
  Week48:Calcium; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Calcium; To High; n=52,45 | 0 | 0
  Week12:Chloride; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Chloride; To Low; n=106,85 | 1 | 2
  Week12:Chloride; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Chloride; To Normal or No Change; n=106,85 | 103 | 82
  Week12:Chloride; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Chloride; To High; n=106,85 | 2 | 1
  Week48:Chloride; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Chloride; To Low; n=52,45 | 1 | 0
  Week48:Chloride; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Chloride; To Normal or No Change; n=52,45 | 51 | 44
  Week48:Chloride; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Chloride; To High; n=52,45 | 0 | 1
  Week12:Creatinine; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Creatinine; To Low; n=106,85 | 0 | 0
  Week12:Creatinine;To Normal or NoChange; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Creatinine;To Normal or NoChange; n=106,85 | 104 | 84
  Week12:Creatinine; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Creatinine; To High; n=106,85 | 2 | 1
  Week48:Creatinine; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Creatinine; To Low; n=52,45 | 3 | 1
  Week48:Creatinine; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Creatinine; To Normal or No Change; n=52,45 | 45 | 42
  Week48:Creatinine; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Creatinine; To High; n=52,45 | 4 | 2
  Week12:Glucose; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Glucose; To Low; n=106,85 | 1 | 2
  Week12:Glucose; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Glucose; To Normal or No Change; n=106,85 | 90 | 72
  Week12:Glucose; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Glucose; To High; n=106,85 | 15 | 11
  Week48:Glucose; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Glucose; To Low; n=52,45 | 0 | 0
  Week48:Glucose; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Glucose; To Normal or No Change; n=52,45 | 44 | 38
  Week48:Glucose; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Glucose; To High; n=52,45 | 8 | 7
  Week12:Potassium; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Potassium; To Low; n=106,85 | 0 | 2
  Week12:Potassium;To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Potassium;To Normal or No Change; n=106,85 | 105 | 83
  Week12:Potassium; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Potassium; To High; n=106,85 | 1 | 0
  Week48:Potassium; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Potassium; To Low; n=52,45 | 0 | 1
  Week48:Potassium; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Potassium; To Normal or No Change; n=52,45 | 52 | 44
  Week48:Potassium; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Potassium; To High; n=52,45 | 0 | 0
  Week12:Sodium; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Sodium; To Low; n=106,85 | 1 | 1
  Week12:Sodium;To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Sodium;To Normal or No Change; n=106,85 | 105 | 84
  Week12:Sodium; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Sodium; To High; n=106,85 | 0 | 0
  Week48:Sodium; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Sodium; To Low; n=52,45 | 2 | 1
  Week48:Sodium;To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Sodium;To Normal or No Change; n=52,45 | 50 | 44
  Week48:Sodium; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Sodium; To High; n=52,45 | 0 | 0
  Week12:T Protein; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:T Protein; To Low; n=106,85 | 10 | 14
  Week12: T Protein;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12: T Protein;To Normal or No Change;n=106,85 | 95 | 71
  Week12:T Protein; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:T Protein; To High; n=106,85 | 1 | 0
  Week48:T Protein; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:T Protein; To Low; n=52,45 | 2 | 3
  Week48:T Protein;To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:T Protein;To Normal or No Change; n=52,45 | 50 | 42
  Week48:T Protein; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:T Protein; To High; n=52,45 | 0 | 0
  Week12:Urea/BUN; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Urea/BUN; To Low; n=106,85 | 2 | 2
  Week12Urea/BUN; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12Urea/BUN; To Normal or No Change; n=106,85 | 101 | 78
  Week12:Urea/BUN; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Urea/BUN; To High; n=106,85 | 3 | 5
  Week48:Urea/BUN; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Urea/BUN; To Low; n=52,45 | 2 | 0
  Week48:Urea/BUN; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Urea/BUN; To Normal or No Change; n=52,45 | 47 | 41
  Week48:Urea/BUN; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Urea/BUN; To High; n=52,45 | 3 | 4
  Week12:Uric acid; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Uric acid; To Low; n=106,85 | 2 | 1
  Week12:Uric acid;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Uric acid;To Normal or No Change;n=106,85 | 98 | 83
  Week12:Uric acid; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Uric acid; To High; n=106,85 | 6 | 1
  Week48:Uric acid; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Uric acid; To Low; n=52,45 | 1 | 1
  Week48:Uric acid;To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Uric acid;To Normal or No Change; n=52,45 | 50 | 43
  Week48:Uric acid; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:Uric acid; To High; n=52,45 | 1 | 1

90. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Shift From Baseline Relative to Normal Range in Chemistry Results
Description: as for outcome 89
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week 12:Albumin; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Albumin; To Low; n=53,40 | 1 | 0
  Week12:Albumin; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Albumin; To Normal or No Change; n=53,40 | 52 | 40
  Week12:Albumin; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Albumin; To High; n=53,40 | 0 | 0
  Week 48:Albumin; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Albumin; To Low; n=55,43 | 1 | 2
  Week48:Albumin; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Albumin; To Normal or No Change; n=55,43 | 54 | 41
  Week48:Albumin; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Albumin; To High; n=55,43 | 0 | 0
  Week12:Alk Phosp; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Alk Phosp; To Low; n=53,40 | 0 | 0
  Week12:Alk Phosp;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Alk Phosp;To Normal or No Change;n=53,40 | 49 | 40
  Week12:Alk Phosp; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Alk Phosp; To High; n=53,40 | 4 | 0
  Week48:Alk Phosp; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Alk Phosp; To Low; n=55,43 | 1 | 0
  Week48:Alk Phosp;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Alk Phosp;To Normal or No Change;n=55,43 | 50 | 43
  Week48:Alk Phosp; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Alk Phosp; To High; n=55,43 | 4 | 0
  Week12:ALT;To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:ALT;To Low; n=53,40 | 0 | 0
  Week12:ALT;To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:ALT;To Normal or No Change; n=53,40 | 53 | 40
  Week12:ALT; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:ALT; To High; n=53,40 | 0 | 0
  Week48:ALT;To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:ALT;To Low; n=55,43 | 0 | 0
  Week48:ALT;To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:ALT;To Normal or No Change; n=55,43 | 55 | 43
  Week48:ALT; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:ALT; To High; n=55,43 | 0 | 0
  Week12:AST;To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:AST;To Low; n=53,40 | 0 | 0
  Week12:AST; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:AST; To Normal or No Change; n=53,40 | 53 | 39
  Week12:AST; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:AST; To High; n=53,40 | 0 | 1
  Week48:AST;To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:AST;To Low; n=55,43 | 0 | 0
  Week48:AST; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:AST; To Normal or No Change; n=55,43 | 55 | 42
  Week48:AST; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:AST; To High; n=55,43 | 0 | 1
  Week12:Direct Bil; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Direct Bil; To Low; n=53,40 | 0 | 0
  Week12:Direct Bil;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Direct Bil;To Normal or No Change;n=53,40 | 53 | 40
  Week12:Direct Bil; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Direct Bil; To High; n=53,40 | 0 | 0
  Week48:Direct Bil; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Direct Bil; To Low; n=55,43 | 0 | 0
  Week48:Direct Bil; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Direct Bil; To Normal or No Change; n=55,43 | 54 | 43
  Week48:Direct Bil; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Direct Bil; To High; n=55,43 | 1 | 0
  Week12:Total Bil; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Total Bil; To Low; n=53,40 | 0 | 1
  Week12:Total Bil;To Normal or NoChange; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Total Bil;To Normal or NoChange; n=53,40 | 51 | 39
  Week12:Total Bil; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Total Bil; To High; n=53,40 | 2 | 0
  Week48:Total Bil; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Total Bil; To Low; n=55,43 | 0 | 0
  Week48:Total Bil; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Total Bil; To Normal or No Change; n=55,43 | 54 | 43
  Week48:Total Bil; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Total Bil; To High; n=55,43 | 1 | 0
  Week12:Calcium; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Calcium; To Low; n=53,40 | 2 | 0
  Week12:Calcium; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Calcium; To Normal or No Change; n=53,40 | 51 | 40
  Week12:Calcium; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Calcium; To High; n=53,40 | 0 | 0
  Week48:Calcium; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Calcium; To Low; n=55,43 | 3 | 2
  Week48:Calcium; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Calcium; To Normal or No Change; n=55,43 | 52 | 41
  Week48:Calcium; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Calcium; To High; n=55,43 | 0 | 0
  Week12:Chloride; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Chloride; To Low; n=53,40 | 1 | 0
  Week12:Chloride; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Chloride; To Normal or No Change; n=53,40 | 52 | 40
  Week12:Chloride; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Chloride; To High; n=53,40 | 0 | 0
  Week48:Chloride; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Chloride; To Low; n=55,43 | 1 | 0
  Week48:Chloride; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Chloride; To Normal or No Change; n=55,43 | 53 | 42
  Week48:Chloride; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Chloride; To High; n=55,43 | 1 | 1
  Week12:Creatinine; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Creatinine; To Low; n=53,40 | 2 | 2
  Week12:Creatinine;To Normal or NoChange; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Creatinine;To Normal or NoChange; n=53,40 | 48 | 38
  Week12:Creatinine; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Creatinine; To High; n=53,40 | 3 | 0
  Week48:Creatinine; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Creatinine; To Low; n=55,43 | 2 | 1
  Week48:Creatinine; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Creatinine; To Normal or No Change; n=55,43 | 51 | 42
  Week48:Creatinine; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Creatinine; To High; n=55,43 | 2 | 0
  Week12:Glucose; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Glucose; To Low; n=53,40 | 2 | 0
  Week12:Glucose; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Glucose; To Normal or No Change; n=53,40 | 45 | 32
  Week12:Glucose; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Glucose; To High; n=53,40 | 6 | 8
  Week48:Glucose; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Glucose; To Low; n=55,43 | 1 | 0
  Week48:Glucose; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Glucose; To Normal or No Change; n=55,43 | 44 | 32
  Week48:Glucose; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Glucose; To High; n=55,43 | 10 | 11
  Week12:Potassium; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Potassium; To Low; n=53,40 | 1 | 2
  Week12:Potassium;To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Potassium;To Normal or No Change; n=53,40 | 52 | 38
  Week12:Potassium; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Potassium; To High; n=53,40 | 0 | 0
  Week48:Potassium; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Potassium; To Low; n=55,43 | 1 | 1
  Week48:Potassium; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Potassium; To Normal or No Change; n=55,43 | 54 | 42
  Week48:Potassium; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Potassium; To High; n=55,43 | 0 | 0
  Week12:Sodium; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Sodium; To Low; n=53,40 | 1 | 0
  Week12:Sodium;To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Sodium;To Normal or No Change; n=53,40 | 52 | 40
  Week12:Sodium; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Sodium; To High; n=53,40 | 0 | 0
  Week48:Sodium; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Sodium; To Low; n=55,43 | 0 | 0
  Week48:Sodium;To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Sodium;To Normal or No Change; n=55,43 | 55 | 43
  Week48:Sodium; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Sodium; To High; n=55,43 | 0 | 0
  Week12:T Protein; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:T Protein; To Low; n=53,40 | 3 | 7
  Week12: T Protein;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12: T Protein;To Normal or No Change;n=53,40 | 50 | 33
  Week12:T Protein; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:T Protein; To High; n=53,40 | 0 | 0
  Week48:T Protein; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Protein; To Low; n=55,43 | 4 | 9
  Week48:T Protein;To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Protein;To Normal or No Change; n=55,43 | 51 | 34
  Week48:T Protein; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Protein; To High; n=55,43 | 0 | 0
  Week12:Urea/BUN; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Urea/BUN; To Low; n=53,40 | 0 | 0
  Week12Urea/BUN; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12Urea/BUN; To Normal or No Change; n=53,40 | 49 | 38
  Week12:Urea/BUN; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Urea/BUN; To High; n=53,40 | 4 | 2
  Week48:Urea/BUN; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Urea/BUN; To Low; n=55,43 | 0 | 1
  Week48:Urea/BUN; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Urea/BUN; To Normal or No Change; n=55,43 | 53 | 41
  Week48:Urea/BUN; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Urea/BUN; To High; n=55,43 | 2 | 1
  Week12:Uric acid; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Uric acid; To Low; n=53,40 | 1 | 0
  Week12:Uric acid;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Uric acid;To Normal or No Change;n=53,40 | 49 | 40
  Week12:Uric acid; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Uric acid; To High; n=53,40 | 3 | 0
  Week48:Uric acid; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Uric acid; To Low; n=55,43 | 1 | 1
  Week48:Uric acid;To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Uric acid;To Normal or No Change; n=55,43 | 51 | 42
  Week48:Uric acid; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Uric acid; To High; n=55,43 | 3 | 0

91. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Shift From Baseline Relative to Normal Range in Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; Basophils, Eosinophils (Eosino), Hemoglobin (Hb), Hematocrit (Hct), Lymphocytes (Lympho), Monocytes, Neutrophil Bands (N bands), Total Neutrophils (T neutro), Platelet count (PC), Red Blood Cell (RBC) count, and White Blood Cell count (WBC). Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose on Day 1), Week 12 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: as for outcome 88
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Week12:Basophils;To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Basophils;To Low; n=122, 122 | 0 | 0
  Week12:Basophils;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Basophils;To Normal or No Change;n=122,122 | 122 | 122
  Week12:Basophils; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Basophils; To High; n=122, 122 | 0 | 0
  Week48:Basophils;To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Basophils;To Low; n=16,36 | 0 | 0
  Week48:Basophils;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Basophils;To Normal or No Change;n=16,36 | 16 | 36
  Week48:Basophils; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Basophils; To High; n=16,36 | 0 | 0
  Week12: Eosino; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12: Eosino; To Low; n=122, 122 | 0 | 0
  Week12: Eosino;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12: Eosino;To Normal or No Change;n=122,122 | 120 | 120
  Week 12:Eosino; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Eosino; To High; n=122, 122 | 2 | 2
  Week48: Eosino; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48: Eosino; To Low; n=16,36 | 0 | 0
  Week48: Eosino;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48: Eosino;To Normal or No Change;n=16,36 | 15 | 36
  Week 48:Eosino; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Eosino; To High; n=16,36 | 1 | 0
  Week 12: Hb;To Low;n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12: Hb;To Low;n=122, 123 | 5 | 3
  Week12: Hb; To Normal or No Change; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12: Hb; To Normal or No Change; n=122, 123 | 116 | 117
  Week 12: Hb; To High; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12: Hb; To High; n=122, 123 | 1 | 3
  Week 48: Hb;To Low;n=16,36: number analyzed (Participants) | 16 | 36
  Week 48: Hb;To Low;n=16,36 | 2 | 0
  Week48: Hb; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48: Hb; To Normal or No Change; n=16,36 | 14 | 36
  Week 48: Hb; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48: Hb; To High; n=16,36 | 0 | 0
  Week 12:Hct; To Low; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12:Hct; To Low; n=122, 123 | 1 | 3
  Week12: Hct;To Normal or No Change; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12: Hct;To Normal or No Change; n=122, 123 | 119 | 117
  Week 12:Hct; To High; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12:Hct; To High; n=122, 123 | 2 | 3
  Week 48:Hct; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Hct; To Low; n=16,36 | 0 | 0
  Week48: Hct;To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48: Hct;To Normal or No Change; n=16,36 | 16 | 36
  Week 48:Hct; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Hct; To High; n=16,36 | 0 | 0
  Week 12:Lympho; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Lympho; To Low; n=122, 122 | 0 | 3
  Week12:Lympho; To Normal or No Change; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:Lympho; To Normal or No Change; n=122, 122 | 121 | 115
  Week 12:Lympho; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Lympho; To High; n=122, 122 | 1 | 4
  Week 48:Lympho; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Lympho; To Low; n=16,36 | 0 | 1
  Week48:Lympho; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Lympho; To Normal or No Change; n=16,36 | 16 | 35
  Week 48:Lympho; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Lympho; To High; n=16,36 | 0 | 0
  Week 12:Monocytes; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Monocytes; To Low; n=122, 122 | 1 | 0
  Week12:Monocytes;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:Monocytes;To Normal or No Change;n=122,122 | 120 | 122
  Week 12:Monocytes; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:Monocytes; To High; n=122, 122 | 1 | 0
  Week 48:Monocytes; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:Monocytes; To Low; n=16,36 | 0 | 0
  Week48:Monocytes;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Monocytes;To Normal or No Change;n=16,36 | 16 | 36
  Week48:Monocytes; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:Monocytes; To High; n=16,36 | 0 | 0
  Week 12:N bands; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week 12:N bands; To Low; n=122, 122 | 1 | 1
  Week12:N bands;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:N bands;To Normal or No Change;n=122,122 | 119 | 120
  Week12:N bands; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:N bands; To High; n=122, 122 | 2 | 1
  Week 48:N bands; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:N bands; To Low; n=16,36 | 1 | 0
  Week48:N bands;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:N bands;To Normal or No Change;n=16,36 | 15 | 35
  Week48:N bands; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:N bands; To High; n=16,36 | 0 | 1
  Week12:T Neutro; To Low; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:T Neutro; To Low; n=122, 122 | 2 | 1
  Week12:T Neutro;To Normal or No Change;n=122,122: number analyzed (Participants) | 122 | 122
  Week12:T Neutro;To Normal or No Change;n=122,122 | 120 | 118
  Week12:T Neutro; To High; n=122, 122: number analyzed (Participants) | 122 | 122
  Week12:T Neutro; To High; n=122, 122 | 0 | 3
  Week48:T Neutro; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Neutro; To Low; n=16,36 | 0 | 0
  Week48:T Neutro;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Neutro;To Normal or No Change;n=16,36 | 16 | 33
  Week48:T Neutro; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:T Neutro; To High; n=16,36 | 0 | 3
  Week12:PC; To Low; n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:PC; To Low; n=122, 123 | 4 | 1
  Week 12:PC; To Normal or No Change; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12:PC; To Normal or No Change; n=122, 123 | 116 | 118
  Week12: PC; To High;n=122, 123: number analyzed (Participants) | 122 | 123
  Week12: PC; To High;n=122, 123 | 2 | 4
  Week48:PC; To Low; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:PC; To Low; n=16,36 | 1 | 0
  Week 48:PC; To Normal or No Change; n=16,36: number analyzed (Participants) | 16 | 36
  Week 48:PC; To Normal or No Change; n=16,36 | 15 | 35
  Week48: PC; To High;n=16,36: number analyzed (Participants) | 16 | 36
  Week48: PC; To High;n=16,36 | 0 | 1
  Week12:RBC count; To Low;n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:RBC count; To Low;n=122, 123 | 6 | 7
  Week12:RBC count;To Normal or No Change;n=122,123: number analyzed (Participants) | 122 | 123
  Week12:RBC count;To Normal or No Change;n=122,123 | 114 | 114
  Week12:RBC count;To High;n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:RBC count;To High;n=122, 123 | 2 | 2
  Week48:RBC count; To Low;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:RBC count; To Low;n=16,36 | 1 | 2
  Week48:RBC count;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:RBC count;To Normal or No Change;n=16,36 | 15 | 34
  Week48:RBC count;To High;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:RBC count;To High;n=16,36 | 0 | 0
  Week12:WBC count; To Low;n=122, 123: number analyzed (Participants) | 122 | 123
  Week12:WBC count; To Low;n=122, 123 | 1 | 6
  Week12:WBC count;To Normal or No Change;n=122,123: number analyzed (Participants) | 122 | 123
  Week12:WBC count;To Normal or No Change;n=122,123 | 120 | 116
  Week12:WBC count; To High; n=122,123: number analyzed (Participants) | 122 | 123
  Week12:WBC count; To High; n=122,123 | 1 | 1
  Week48:WBC count; To Low;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:WBC count; To Low;n=16,36 | 1 | 0
  Week48:WBC count;To Normal or No Change;n=16,36: number analyzed (Participants) | 16 | 36
  Week48:WBC count;To Normal or No Change;n=16,36 | 15 | 35
  Week48:WBC count; To High; n=16,36: number analyzed (Participants) | 16 | 36
  Week48:WBC count; To High; n=16,36 | 0 | 1

92. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Shift From Baseline Relative to Normal Range in Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; Basophils, Eosino, Hb, Hct, Lympho, Monocytes, N bands, T neutro, PC, RBC count, and WBC. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: as for outcome 89
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week12:Basophils;To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Basophils;To Low; n=106,85 | 0 | 0
  Week12:Basophils;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Basophils;To Normal or No Change;n=106,85 | 106 | 85
  Week12:Basophils; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Basophils; To High; n=106,85 | 0 | 0
  Week48:Basophils;To Low; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Basophils;To Low; n=52,44 | 0 | 0
  Week48:Basophils;To Normal or No Change;n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Basophils;To Normal or No Change;n=52,44 | 52 | 44
  Week48:Basophils; To High; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Basophils; To High; n=52,44 | 0 | 0
  Week12: Eosino; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12: Eosino; To Low; n=106,85 | 0 | 0
  Week12: Eosino;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12: Eosino;To Normal or No Change;n=106,85 | 105 | 85
  Week 12:Eosino; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Eosino; To High; n=106,85 | 1 | 0
  Week48: Eosino; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48: Eosino; To Low; n=52,45 | 0 | 0
  Week48: Eosino;To Normal or No Change;n=52,45: number analyzed (Participants) | 52 | 45
  Week48: Eosino;To Normal or No Change;n=52,45 | 51 | 43
  Week 48:Eosino; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48:Eosino; To High; n=52,45 | 1 | 1
  Week 12: Hb;To Low;n=106,85: number analyzed (Participants) | 106 | 85
  Week 12: Hb;To Low;n=106,85 | 4 | 3
  Week12: Hb; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12: Hb; To Normal or No Change; n=106,85 | 101 | 81
  Week 12: Hb; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12: Hb; To High; n=106,85 | 1 | 1
  Week 48: Hb;To Low;n=52,45: number analyzed (Participants) | 52 | 45
  Week 48: Hb;To Low;n=52,45 | 3 | 3
  Week48: Hb; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48: Hb; To Normal or No Change; n=52,45 | 49 | 41
  Week 48: Hb; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48: Hb; To High; n=52,45 | 0 | 1
  Week 12:Hct; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Hct; To Low; n=106,85 | 3 | 1
  Week12: Hct;To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12: Hct;To Normal or No Change; n=106,85 | 100 | 80
  Week 12:Hct; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Hct; To High; n=106,85 | 3 | 4
  Week 48:Hct; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48:Hct; To Low; n=52,45 | 1 | 1
  Week48: Hct;To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week48: Hct;To Normal or No Change; n=52,45 | 48 | 43
  Week 48:Hct; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48:Hct; To High; n=52,45 | 3 | 1
  Week 12:Lympho; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Lympho; To Low; n=106,85 | 0 | 1
  Week12:Lympho; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Lympho; To Normal or No Change; n=106,85 | 101 | 83
  Week 12:Lympho; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Lympho; To High; n=106,85 | 5 | 1
  Week 48:Lympho; To Low; n=52,44: number analyzed (Participants) | 52 | 44
  Week 48:Lympho; To Low; n=52,44 | 2 | 2
  Week48:Lympho; To Normal or No Change; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Lympho; To Normal or No Change; n=52,44 | 49 | 40
  Week 48:Lympho; To High; n=52,44: number analyzed (Participants) | 52 | 44
  Week 48:Lympho; To High; n=52,44 | 1 | 2
  Week 12:Monocytes; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Monocytes; To Low; n=106,85 | 1 | 1
  Week12:Monocytes;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:Monocytes;To Normal or No Change;n=106,85 | 105 | 83
  Week 12:Monocytes; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:Monocytes; To High; n=106,85 | 0 | 1
  Week 48:Monocytes; To Low; n=52,44: number analyzed (Participants) | 52 | 44
  Week 48:Monocytes; To Low; n=52,44 | 0 | 0
  Week48:Monocytes;To Normal or No Change;n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Monocytes;To Normal or No Change;n=52,44 | 52 | 44
  Week48:Monocytes; To High; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:Monocytes; To High; n=52,44 | 0 | 0
  Week 12:N bands; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:N bands; To Low; n=106,85 | 2 | 1
  Week12:N bands;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:N bands;To Normal or No Change;n=106,85 | 104 | 83
  Week12:N bands; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:N bands; To High; n=106,85 | 0 | 1
  Week 48:N bands; To Low; n=52,44: number analyzed (Participants) | 52 | 44
  Week 48:N bands; To Low; n=52,44 | 0 | 1
  Week48:N bands;To Normal or No Change;n=52,44: number analyzed (Participants) | 52 | 44
  Week48:N bands;To Normal or No Change;n=52,44 | 52 | 43
  Week48:N bands; To High; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:N bands; To High; n=52,44 | 0 | 0
  Week12:T Neutro; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:T Neutro; To Low; n=106,85 | 3 | 1
  Week12:T Neutro;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:T Neutro;To Normal or No Change;n=106,85 | 103 | 82
  Week12:T Neutro; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:T Neutro; To High; n=106,85 | 0 | 2
  Week48:T Neutro; To Low; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:T Neutro; To Low; n=52,44 | 0 | 2
  Week48:T Neutro;To Normal or No Change;n=52,44: number analyzed (Participants) | 52 | 44
  Week48:T Neutro;To Normal or No Change;n=52,44 | 50 | 41
  Week48:T Neutro; To High; n=52,44: number analyzed (Participants) | 52 | 44
  Week48:T Neutro; To High; n=52,44 | 2 | 1
  Week12:PC; To Low; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:PC; To Low; n=106,85 | 0 | 0
  Week 12:PC; To Normal or No Change; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12:PC; To Normal or No Change; n=106,85 | 105 | 83
  Week12: PC; To High;n=106,85: number analyzed (Participants) | 106 | 85
  Week12: PC; To High;n=106,85 | 1 | 2
  Week48:PC; To Low; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:PC; To Low; n=52,45 | 0 | 0
  Week 48:PC; To Normal or No Change; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48:PC; To Normal or No Change; n=52,45 | 51 | 45
  Week48: PC; To High;n=52,45: number analyzed (Participants) | 52 | 45
  Week48: PC; To High;n=52,45 | 1 | 0
  Week12:RBC count; To Low;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:RBC count; To Low;n=106,85 | 5 | 3
  Week12:RBC count;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:RBC count;To Normal or No Change;n=106,85 | 98 | 80
  Week12:RBC count;To High;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:RBC count;To High;n=106,85 | 3 | 2
  Week48:RBC count; To Low;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:RBC count; To Low;n=52,45 | 5 | 1
  Week48:RBC count;To Normal or No Change;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:RBC count;To Normal or No Change;n=52,45 | 47 | 44
  Week48:RBC count;To High;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:RBC count;To High;n=52,45 | 0 | 0
  Week12:WBC count; To Low;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:WBC count; To Low;n=106,85 | 0 | 1
  Week12:WBC count;To Normal or No Change;n=106,85: number analyzed (Participants) | 106 | 85
  Week12:WBC count;To Normal or No Change;n=106,85 | 106 | 82
  Week12:WBC count; To High; n=106,85: number analyzed (Participants) | 106 | 85
  Week12:WBC count; To High; n=106,85 | 0 | 2
  Week48:WBC count; To Low;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:WBC count; To Low;n=52,45 | 0 | 3
  Week48:WBC count;To Normal or No Change;n=52,45: number analyzed (Participants) | 52 | 45
  Week48:WBC count;To Normal or No Change;n=52,45 | 52 | 41
  Week48:WBC count; To High; n=52,45: number analyzed (Participants) | 52 | 45
  Week48:WBC count; To High; n=52,45 | 0 | 1

93. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Shift From Baseline Relative to Normal Range in Hematology Parameters
Description: as for outcome 92
Time Frame: as for outcome 90
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week12:Basophils;To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Basophils;To Low; n=53,40 | 0 | 0
  Week12:Basophils;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Basophils;To Normal or No Change;n=53,40 | 53 | 40
  Week12:Basophils; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Basophils; To High; n=53,40 | 0 | 0
  Week48:Basophils;To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Basophils;To Low; n=55,43 | 0 | 0
  Week48:Basophils;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Basophils;To Normal or No Change;n=55,43 | 55 | 43
  Week48:Basophils; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Basophils; To High; n=55,43 | 0 | 0
  Week12: Eosino; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12: Eosino; To Low; n=53,40 | 0 | 0
  Week12: Eosino;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12: Eosino;To Normal or No Change;n=53,40 | 52 | 38
  Week 12:Eosino; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Eosino; To High; n=53,40 | 1 | 2
  Week48: Eosino; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48: Eosino; To Low; n=55,43 | 0 | 0
  Week48: Eosino;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48: Eosino;To Normal or No Change;n=55,43 | 54 | 41
  Week 48:Eosino; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Eosino; To High; n=55,43 | 1 | 2
  Week 12: Hb;To Low;n=53,40: number analyzed (Participants) | 53 | 40
  Week 12: Hb;To Low;n=53,40 | 1 | 0
  Week12: Hb; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12: Hb; To Normal or No Change; n=53,40 | 51 | 40
  Week 12: Hb; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12: Hb; To High; n=53,40 | 1 | 0
  Week 48: Hb;To Low;n=55,43: number analyzed (Participants) | 55 | 43
  Week 48: Hb;To Low;n=55,43 | 0 | 2
  Week48: Hb; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48: Hb; To Normal or No Change; n=55,43 | 54 | 39
  Week 48: Hb; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48: Hb; To High; n=55,43 | 1 | 2
  Week 12:Hct; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Hct; To Low; n=53,40 | 1 | 0
  Week12: Hct;To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12: Hct;To Normal or No Change; n=53,40 | 51 | 38
  Week 12:Hct; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Hct; To High; n=53,40 | 1 | 2
  Week 48:Hct; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Hct; To Low; n=55,43 | 0 | 1
  Week48: Hct;To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48: Hct;To Normal or No Change; n=55,43 | 53 | 41
  Week 48:Hct; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Hct; To High; n=55,43 | 2 | 1
  Week 12:Lympho; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Lympho; To Low; n=53,40 | 0 | 1
  Week12:Lympho; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Lympho; To Normal or No Change; n=53,40 | 53 | 39
  Week 12:Lympho; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Lympho; To High; n=53,40 | 0 | 0
  Week 48:Lympho; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Lympho; To Low; n=55,43 | 2 | 1
  Week48:Lympho; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Lympho; To Normal or No Change; n=55,43 | 51 | 41
  Week 48:Lympho; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Lympho; To High; n=55,43 | 2 | 1
  Week 12:Monocytes; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Monocytes; To Low; n=53,40 | 0 | 0
  Week12:Monocytes;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:Monocytes;To Normal or No Change;n=53,40 | 53 | 40
  Week 12:Monocytes; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:Monocytes; To High; n=53,40 | 0 | 0
  Week 48:Monocytes; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:Monocytes; To Low; n=55,43 | 0 | 0
  Week48:Monocytes;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Monocytes;To Normal or No Change;n=55,43 | 54 | 43
  Week48:Monocytes; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:Monocytes; To High; n=55,43 | 1 | 0
  Week 12:N bands; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:N bands; To Low; n=53,40 | 1 | 0
  Week12:N bands;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:N bands;To Normal or No Change;n=53,40 | 50 | 40
  Week12:N bands; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:N bands; To High; n=53,40 | 2 | 0
  Week 48:N bands; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:N bands; To Low; n=55,43 | 1 | 0
  Week48:N bands;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:N bands;To Normal or No Change;n=55,43 | 52 | 43
  Week48:N bands; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:N bands; To High; n=55,43 | 2 | 0
  Week12:T Neutro; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:T Neutro; To Low; n=53,40 | 0 | 1
  Week12:T Neutro;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:T Neutro;To Normal or No Change;n=53,40 | 53 | 38
  Week12:T Neutro; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:T Neutro; To High; n=53,40 | 0 | 1
  Week48:T Neutro; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Neutro; To Low; n=55,43 | 2 | 1
  Week48:T Neutro;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Neutro;To Normal or No Change;n=55,43 | 52 | 39
  Week48:T Neutro; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:T Neutro; To High; n=55,43 | 1 | 3
  Week12:PC; To Low; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:PC; To Low; n=53,40 | 0 | 0
  Week 12:PC; To Normal or No Change; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12:PC; To Normal or No Change; n=53,40 | 52 | 40
  Week12: PC; To High;n=53,40: number analyzed (Participants) | 53 | 40
  Week12: PC; To High;n=53,40 | 1 | 0
  Week48:PC; To Low; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:PC; To Low; n=55,43 | 0 | 0
  Week 48:PC; To Normal or No Change; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48:PC; To Normal or No Change; n=55,43 | 54 | 42
  Week48: PC; To High;n=55,43: number analyzed (Participants) | 55 | 43
  Week48: PC; To High;n=55,43 | 1 | 1
  Week12:RBC count; To Low;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:RBC count; To Low;n=53,40 | 2 | 2
  Week12:RBC count;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:RBC count;To Normal or No Change;n=53,40 | 51 | 38
  Week12:RBC count;To High;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:RBC count;To High;n=53,40 | 0 | 0
  Week48:RBC count; To Low;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:RBC count; To Low;n=55,43 | 1 | 4
  Week48:RBC count;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:RBC count;To Normal or No Change;n=55,43 | 54 | 37
  Week48:RBC count;To High;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:RBC count;To High;n=55,43 | 0 | 2
  Week12:WBC count; To Low;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:WBC count; To Low;n=53,40 | 1 | 0
  Week12:WBC count;To Normal or No Change;n=53,40: number analyzed (Participants) | 53 | 40
  Week12:WBC count;To Normal or No Change;n=53,40 | 50 | 40
  Week12:WBC count; To High; n=53,40: number analyzed (Participants) | 53 | 40
  Week12:WBC count; To High; n=53,40 | 2 | 0
  Week48:WBC count; To Low;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:WBC count; To Low;n=55,43 | 3 | 1
  Week48:WBC count;To Normal or No Change;n=55,43: number analyzed (Participants) | 55 | 43
  Week48:WBC count;To Normal or No Change;n=55,43 | 51 | 42
  Week48:WBC count; To High; n=55,43: number analyzed (Participants) | 55 | 43
  Week48:WBC count; To High; n=55,43 | 1 | 0

94. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Worst Case Post-Baseline Urinalysis Results Relative to Baseline
Description: Urine samples were collected for analysis of presence of occult blood and protein in urine using dipstick method. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of occult blood and protein can be read as negative, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations in the urine sample. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose on Day 1) and up to 48 weeks in Treatment Cycle 1
Population: SPDB Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Occult Blood; No Change/Decreased | 98 | 92
  Occult Blood; Any Increase | 26 | 32
  Occult Blood; Increase to Traces | 7 | 11
  Occult Blood; Increase to 1+ | 14 | 8
  Occult Blood; Increase to 2+ | 4 | 7
  Occult Blood; Increase to 3+ | 1 | 6
  Occult Blood; Increase to 4+ | 0 | 0
  Protein; No Change/Decreased | 105 | 111
  Protein; Any Increase | 19 | 13
  Protein; Increase to Traces | 7 | 5
  Protein; Increase to 1+ | 9 | 7
  Protein; Increase to 2+ | 3 | 1
  Protein; Increase to 3+ | 0 | 0
  Protein; Increase to 4+ | 0 | 0

95. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Worst Case Post-Baseline Urinalysis Results Relative to Baseline
Description: as for outcome 94
Time Frame: Baseline (Pre-dose of Treatment Cycle 1) and up to 48 weeks after 1st treatment
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Occult Blood; No Change/Decreased, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; No Change/Decreased, n=108,88 | 70 | 54
  Occult Blood; Any Increase, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Any Increase, n=108,88 | 38 | 34
  Occult Blood; Increase to Traces, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Increase to Traces, n=108,88 | 12 | 10
  Occult Blood; Increase to 1+, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Increase to 1+, n=108,88 | 11 | 10
  Occult Blood; Increase to 2+, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Increase to 2+, n=108,88 | 11 | 7
  Occult Blood; Increase to 3+, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Increase to 3+, n=108,88 | 4 | 7
  Occult Blood; Increase to 4+, n=108,88: number analyzed (Participants) | 108 | 88
  Occult Blood; Increase to 4+, n=108,88 | 0 | 0
  Protein;No Change/Decreased, n=108,88: number analyzed (Participants) | 108 | 88
  Protein;No Change/Decreased, n=108,88 | 80 | 72
  Protein;Any Increase, n=108,88: number analyzed (Participants) | 108 | 88
  Protein;Any Increase, n=108,88 | 28 | 16
  Protein; Increase to Traces, n=108,88: number analyzed (Participants) | 108 | 88
  Protein; Increase to Traces, n=108,88 | 14 | 7
  Protein; Increase to 1+, n=108,88: number analyzed (Participants) | 108 | 88
  Protein; Increase to 1+, n=108,88 | 8 | 8
  Protein; Increase to 2+, n=108,88: number analyzed (Participants) | 108 | 88
  Protein; Increase to 2+, n=108,88 | 4 | 1
  Protein; Increase to 3+, n=108,88: number analyzed (Participants) | 108 | 88
  Protein; Increase to 3+, n=108,88 | 2 | 0
  Protein; Increase to 4+, n=108,88: number analyzed (Participants) | 108 | 88
  Protein; Increase to 4+, n=108,88 | 0 | 0

96. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Worst Case Post-Baseline Urinalysis Results Relative to Baseline
Description: as for outcome 94
Time Frame: Baseline (Pre-dose of Treatment Cycle 1) and up to 48 weeks after 1st treatment
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Occult Blood; No Change/Decreased, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; No Change/Decreased, n=56,43 | 40 | 25
  Occult Blood; Any Increase, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Any Increase, n=56,43 | 16 | 18
  Occult Blood; Increase to Traces, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Increase to Traces, n=56,43 | 3 | 3
  Occult Blood; Increase to 1+, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Increase to 1+, n=56,43 | 5 | 8
  Occult Blood; Increase to 2+, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Increase to 2+, n=56,43 | 5 | 3
  Occult Blood; Increase to 3+, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Increase to 3+, n=56,43 | 3 | 4
  Occult Blood; Increase to 4+, n=56,43: number analyzed (Participants) | 56 | 43
  Occult Blood; Increase to 4+, n=56,43 | 0 | 0
  Protein;No Change/Decreased, n=56,43: number analyzed (Participants) | 56 | 43
  Protein;No Change/Decreased, n=56,43 | 44 | 37
  Protein;Any Increase, n=56,43: number analyzed (Participants) | 56 | 43
  Protein;Any Increase, n=56,43 | 12 | 6
  Protein; Increase to Traces, n=56,43: number analyzed (Participants) | 56 | 43
  Protein; Increase to Traces, n=56,43 | 3 | 4
  Protein; Increase to 1+, n=56,43: number analyzed (Participants) | 56 | 43
  Protein; Increase to 1+, n=56,43 | 4 | 2
  Protein; Increase to 2+, n=56,43: number analyzed (Participants) | 56 | 43
  Protein; Increase to 2+, n=56,43 | 5 | 0
  Protein; Increase to 3+, n=56,43: number analyzed (Participants) | 56 | 43
  Protein; Increase to 3+, n=56,43 | 0 | 0
  Protein; Increase to 4+, n=56,43: number analyzed (Participants) | 56 | 43
  Protein; Increase to 4+, n=56,43 | 0 | 0

97. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Urinary Tract Infection (UTI)
Description: A urine culture and sensitivity test were performed when urinalysis results with a urine reagent strip are suggestive of a UTI (positive nitrites or leukocyte esterase). UTI was recorded as an AE, irrespective of symptoms when the result of urine culture was positive (with the presence of bacteriuria with >=10^5 Colony Forming Unit per milliliter (CFU/mL) and leukocyturia with >5 per high power field was noted.
Time Frame: Up to 48 weeks in Treatment Cycle 1
Population: SPDB Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants | 10 | 22

98. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With UTI: Placebo/GSK1358820 100 U
Description: A urine culture and sensitivity test were performed when urinalysis results with a urine reagent strip are suggestive of a UTI (positive nitrites or leukocyte esterase). UTI was recorded as an AE, irrespective of symptoms when the result of urine culture was positive (with the presence of bacteriuria with >=10^5 CFU/mL and leukocyturia with >5 per high power field was noted.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Participants | 30

99. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With UTI: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 98
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 88
Participants | 19

100. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With UTI: Placebo/GSK1358820 100 U
Description: as for outcome 98
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 56
Participants | 15

101. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With UTI: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 98
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 43
Participants | 14

102. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Change From Baseline in PVR Urine Volume
Description: PVR urine volume was assessed by ultrasound or bladder scan after participants perform a voluntary void according to the study schedule. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as any visit value minus Baseline value.
Time Frame: as for outcome 73
Population: as for outcome 88
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Milliliter
  Week 2; n=124, 123: number analyzed (Participants) | 124 | 123
  Week 2; n=124, 123 | 1.02 (28.801) | 44.99 (76.009)
  Week 6; n=124, 122: number analyzed (Participants) | 124 | 122
  Week 6; n=124, 122 | 1.42 (36.387) | 25.62 (50.820)
  Week 12; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; n=122, 123 | 4.05 (39.432) | 16.81 (35.717)
  Week 18; n=23, 65: number analyzed (Participants) | 23 | 65
  Week 18; n=23, 65 | 8.91 (52.093) | 16.10 (42.109)
  Week 24; n=17, 54: number analyzed (Participants) | 17 | 54
  Week 24; n=17, 54 | 2.92 (37.846) | 18.06 (45.829)
  Week 30; n=14, 47: number analyzed (Participants) | 14 | 47
  Week 30; n=14, 47 | 19.96 (78.149) | 13.33 (39.357)
  Week 36; n=12, 32: number analyzed (Participants) | 12 | 32
  Week 36; n=12, 32 | 2.25 (35.433) | 9.87 (36.672)
  Week 42; n=11, 27: number analyzed (Participants) | 11 | 27
  Week 42; n=11, 27 | -15.26 (42.147) | 10.83 (38.952)
  Week 48; n=16, 36: number analyzed (Participants) | 16 | 36
  Week 48; n=16, 36 | 10.93 (69.151) | 5.56 (35.878)

103. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in PVR Urine Volume: Placebo/GSK1358820 100 U
Description: as for outcome 102
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Milliliter
  Week 2; n=108 | 34.87 (56.255)
  Week 6; n=108 | 30.11 (53.625)
  Week 12; n=106: number analyzed (Participants) | 106
  Week 12; n=106 | 19.33 (40.498)
  Week 18; n=82: number analyzed (Participants) | 82
  Week 18; n=82 | 15.09 (46.604)
  Week 24; n=45: number analyzed (Participants) | 45
  Week 24; n=45 | 19.11 (40.219)
  Week 30; n=37: number analyzed (Participants) | 37
  Week 30; n=37 | 5.66 (29.172)
  Week 36; n=7: number analyzed (Participants) | 7
  Week 36; n=7 | 3.69 (28.760)
  Week 48; n=52: number analyzed (Participants) | 52
  Week 48; n=52 | 10.98 (40.499)

104. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in PVR Urine Volume: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 102
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 2, Week 6, Week 12, Week 18, Week 24, Week 30 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Milliliter
  Week 2; n=86: number analyzed (Participants) | 86
  Week 2; n=86 | 36.72 (54.171)
  Week 6; n=86: number analyzed (Participants) | 86
  Week 6; n=86 | 30.26 (43.818)
  Week 12; n=85: number analyzed (Participants) | 85
  Week 12; n=85 | 17.06 (42.424)
  Week 18; n=39: number analyzed (Participants) | 39
  Week 18; n=39 | 20.15 (48.934)
  Week 24; n=19: number analyzed (Participants) | 19
  Week 24; n=19 | 5.38 (25.570)
  Week 30; n=14: number analyzed (Participants) | 14
  Week 30; n=14 | 18.61 (31.086)
  Week 48; n=45: number analyzed (Participants) | 45
  Week 48; n=45 | 12.18 (46.394)

105. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in PVR Urine Volume: Placebo/GSK1358820 100 U
Description: as for outcome 102
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 2, Week 6, Week 12, Week 18, Week 24 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Milliliter
  Week 2; n=56: number analyzed (Participants) | 56
  Week 2; n=56 | 49.97 (64.295)
  Week 6; n=55: number analyzed (Participants) | 55
  Week 6; n=55 | 36.32 (49.891)
  Week 12; n=53: number analyzed (Participants) | 53
  Week 12; n=53 | 25.20 (49.651)
  Week 18; n=19: number analyzed (Participants) | 19
  Week 18; n=19 | 32.57 (59.514)
  Week 24; n=1: number analyzed (Participants) | 1
  Week 24; n=1 | 39.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 48; n=56: number analyzed (Participants) | 56
  Week 48; n=56 | 26.65 (54.171)

106. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in PVR Urine Volume: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 102
Time Frame: Baseline (Pre-dose of Treatment Cycle 1), Week 2, Week 6, Week 12, Week 18 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: as for outcome 75
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 124
Milliliter
  Week 2; n=43: number analyzed (Participants) | 43
  Week 2; n=43 | 50.13 (59.960)
  Week 6; n=43: number analyzed (Participants) | 43
  Week 6; n=43 | 28.09 (42.401)
  Week 12; n=40: number analyzed (Participants) | 40
  Week 12; n=40 | 24.96 (42.308)
  Week 18; n=27: number analyzed (Participants) | 27
  Week 18; n=27 | 14.54 (42.237)
  Week 48; n=43: number analyzed (Participants) | 43
  Week 48; n=43 | 22.85 (48.338)

107. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants Using Clean Intermittent Catheterization (CIC) for Urinary Retention or Elevated PVR
Description: Participants who had used CIC at least once after the first treatment with the reason for urinary retention or elevated PVR have been presented.
Time Frame: Up to 48 weeks in Treatment Cycle 1
Population: SPDB Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants | 2 | 7

108. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: Placebo/GSK1358820 100 U
Description: as for outcome 107
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Participants | 3

109. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 107
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 88
Participants | 3

110. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: Placebo/GSK1358820 100 U
Description: as for outcome 107
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 56
Participants | 2

111. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 107
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 43
Participants | 0

112. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Abnormal Findings Undergoing Kidney and Bladder Ultrasound
Description: The kidney and bladder ultrasound was performed in order to assess the presence of stones in the kidneys and bladder, an ultrasound of these structures (with the bladder at least half full) was performed. Participants with abnormal findings after kidney and bladder ultrasound have been presented.
Time Frame: Up to 48 weeks in Treatment Cycle 1
Population: SPDB Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Kidney ultrasound | 3 | 4
  Bladder ultrasound | 0 | 0

113. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Abnormal Findings Undergoing Kidney and Bladder Ultrasound: Placebo/GSK1358820 100 U
Description: as for outcome 112
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 108
Participants
  Kidney ultrasound | 2
  Bladder ultrasound | 0

114. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Abnormal Findings Undergoing Kidney and Bladder Ultrasound: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 112
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 88
Participants
  Kidney ultrasound | 2
  Bladder ultrasound | 0

115. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Abnormal Findings Undergoing Kidney and Bladder Ultrasound: Placebo/GSK1358820 100 U
Description: as for outcome 112
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U
Number analyzed (Participants) | 56
Participants
  Kidney ultrasound | 1
  Bladder ultrasound | 0

116. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Abnormal Findings Undergoing Kidney and Bladder Ultrasound: GSK1358820 100 U/GSK1358820 100 U
Description: as for outcome 112
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 43
Participants
  Kidney ultrasound | 0
  Bladder ultrasound | 0

117. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1): Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single 12-lead ECGs were obtained at indicated time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS and QT interval. QT interval corrected for heart rate (QTc) value is machine-read or manually over-read. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Baseline (Pre-dose on Day 1), Week 12 and Week 48 in Treatment Cycle 1
Population: as for outcome 73
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U
Number analyzed (Participants) | 124 | 124
Participants
  Baseline; NCS; n=124, 124 | 25 | 31
  Baseline; CS; n=124, 124 | 3 | 1
  Week 12; NCS; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; NCS; n=122, 123 | 28 | 28
  Week 12; CS; n=122, 123: number analyzed (Participants) | 122 | 123
  Week 12; CS; n=122, 123 | 1 | 1
  Week 48; NCS; n=16, 36: number analyzed (Participants) | 16 | 36
  Week 48; NCS; n=16, 36 | 1 | 6
  Week 48; CS; n=16, 36: number analyzed (Participants) | 16 | 36
  Week 48; CS; n=16, 36 | 0 | 0

118. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Abnormal ECG Findings
Description: Single 12-lead ECGs were obtained at indicated time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS and QT interval. QTc value is machine-read or manually over-read. CS and NCS abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week 12; NCS; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; NCS; n=106,85 | 29 | 25
  Week 12; CS; n=106,85: number analyzed (Participants) | 106 | 85
  Week 12; CS; n=106,85 | 0 | 0
  Week 48; NCS; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48; NCS; n=52,45 | 11 | 13
  Week 48; CS; n=52,45: number analyzed (Participants) | 52 | 45
  Week 48; CS; n=52,45 | 1 | 0

119. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Abnormal ECG Findings
Description: as for outcome 118
Time Frame: Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
Number analyzed (Participants) | 108 | 124
Participants
  Week 12; NCS; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12; NCS; n=53,40 | 10 | 9
  Week 12; CS; n=53,40: number analyzed (Participants) | 53 | 40
  Week 12; CS; n=53,40 | 0 | 0
  Week 48; NCS; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48; NCS; n=55,43 | 17 | 12
  Week 48; CS; n=55,43: number analyzed (Participants) | 55 | 43
  Week 48; CS; n=55,43 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and Non-SAEs were collected from start of the first treatment up to 48 weeks in Treatment Cycle 1 and up to Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycles 2 and 3
Description: SAEs and non-SAEs were reported for SPDB Population (Treatment Cycle1:Placebo and GSK1358820 100 U) and Safety Populations 1 (Treatment Cycle2:Placebo/GSK1358820 100 U), 2 (Treatment Cycle 2:GSK1358820 100 U/GSK1358820 100 U and Treatment Cycle 3: Placebo/GSK1358820 100 U) and 3 (Treatment Cycle3:GSK1358820 100 U/GSK1358820 100 U).
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 100 U | Treatment Cycle 2: Placebo / GSK1358820 100 U | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U | Treatment Cycle 3: Placebo / GSK1358820 100 U | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124 | 0/108 | 0/88 | 0/56 | 0/43
Serious Adverse Events (participants affected / at risk) | 6/124 | 8/124 | 5/108 | 5/88 | 0/56 | 1/43
Other Adverse Events (participants affected / at risk) | 29/124 | 53/124 | 49/108 | 40/88 | 22/56 | 19/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Cycle 1: Placebo (N=124) | Treatment Cycle 1: GSK1358820 100 U (N=124) | Treatment Cycle 2: Placebo / GSK1358820 100 U (N=108) | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U (N=88) | Treatment Cycle 3: Placebo / GSK1358820 100 U (N=56) | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U (N=43)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Cycle 1: Placebo (N=124) | Treatment Cycle 1: GSK1358820 100 U (N=124) | Treatment Cycle 2: Placebo / GSK1358820 100 U (N=108) | Treatment Cycle 2: GSK1358820 100 U / GSK1358820 100 U (N=88) | Treatment Cycle 3: Placebo / GSK1358820 100 U (N=56) | Treatment Cycle 3: GSK1358820 100 U / GSK1358820 100 U (N=43)
Nasopharyngitis (Infections and infestations) | 13 (14) | 22 (26) | 14 (18) | 14 (14) | 5 (8) | 5 (6)
Urinary tract infection (Infections and infestations) | 10 (11) | 22 (31) | 30 (40) | 19 (22) | 15 (19) | 14 (17)
Cystitis (Infections and infestations) | 2 (2) | 9 (9) | 4 (5) | 5 (5) | 9 (13) | 3 (3)
Dysuria (Renal and urinary disorders) | 3 (4) | 14 (15) | 4 (4) | 5 (5) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Residual urine volume increased (Investigations) | 0 (0) | 7 (7) | 3 (3) | 6 (6) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT02820844/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02820844/SAP_001.pdf